| | | CLIN-PROT-CIP-11-050069 |
|---------------|------------------------|-------------------------|
| 31 <b>V</b> 1 | CLINICAL INVESTIGATION | Version: 3 |
| HealthCare | PLAN | Status: Release |

| Study Title | Prospective, randomized, split-mouth study evaluating the clinical performance of a new dental adhesive, $3M^{TM}$ Scotchbond <sup>TM</sup> Universal Plus Adhesive, compared to $3M^{TM}$ Scotchbond <sup>TM</sup> Universal Adhesive when used for posterior Class I and Class II restorations with $3M^{TM}$ Filtek <sup>TM</sup> Universal Restorative |
|---|---|
| Study Number | EM-11-050069 |
| CIP Version | 1 |
| Release Date | 01/27/2022 08:22:29 AM CST |
| Name of Device<br>Under Investigation | Scotchbond <sup>TM</sup> Universal Plus |
| Sponsor Address | 3M Company 3M Healthcare Business Group 3M Center – 270-4N St. Paul, MN. 55144 |
| Manufacturer<br>Address | 3M Deutschland GmbH<br>Carl-Schurz-Str. 1<br>41453 Neuss -Germany |

#### **ELECTRONIC SIGNATURES:**

| Signer | Role | Date Signed |
|---|---|---|
| us267473:Myhre Paula E | Clinical | January 27, 2022 08:22:09 AM CST |
| GES10885:Wittig-Barger Ulrice | Regulatory and | January 27, 2022 04:22:04 AM CST |
| GES10883. Wittig-Barger Office | Compliance | January 27, 2022 04.22.04 AM CS1 |
| AASAAZZ:Lin Chee Paul | Clinical | January 26, 2022 11:33:54 AM CST |
| ge320710:Syrek Andreas | Medical Monitor | January 27, 2022 01:42:53 AM CST |

#### 3M Confidential

This document contains confidential information that is the property of 3M and is subject to all the restrictions on its use and disclosure contained in the study contract to which this is appended. Do not copy, disclose, circulate, or use for benefit for any third party without written authorization from 3M.

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 

## CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069

Version: 3 Status: Release

#### **Investigator Statements of Compliance**

This clinical investigation shall be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki.

This clinical investigation shall be conducted in accordance with ISO-14155:2011 and future versions, US FDA 21 CFR parts 812, 50, 54, 56, and any regional or national regulations, as appropriate.

The clinical investigation shall not begin until the required approval/favorable opinion from the Institutional Review Board (IRB)/Ethics Committee (EC) and regulatory authority (if applicable) has been obtained and permission to proceed has been received from the study Sponsor. Any additional requirements imposed by the IRB/EC or regulatory authority shall be followed.

I have read the Clinical Investigation Plan (CIP), including all appendices, as well as supporting study related documents and I agree that it contains all necessary details for me and my staff to conduct this study as described. I agree to record all adverse events/ deviations and report those adverse events/ deviations to the Sponsor per this CIP and IRB/EC per local requirements. I always agree to maintain product accountability and ensure security of study materials. I agree to comply with financial disclosure requirements.

All subjects will sign and date the approved Informed Consent before any study procedures are conducted, as applicable

I will ensure that all subjects meet inclusion criteria before enrolling them in the study.

I agree to maintain and retain records as required by this Clinical Investigation Plan.

| Investigator's Signature: | | Date: |
|---|---|---|
| Investigator's Name: | Jorge Perdigao, DMD, MS, PhD | |
| Institution: | University of Minnesota School of Dentistry Department of Restorative Sciences | |
| Investigator's<br>Signature: | | Date: |
| Investigator's Name: | Hooi Pin Chew (BDS, FDSRCS, PhD) | |
| Institution: | University of Minnesota School of Dentistry Department of Restorative Sciences | |

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


#### ABBREVIATIONS/ACRONYMS

| ADE | adverse device effect |
|-------|--------------------------------------------------------------|
| AE | adverse event |
| AFR | annual fail rate |
| ASA | American Society for Anesthesiologists |
| BPA | bisphenol A |
| CIP | Clinical Investigation Plan |
| Co-PI | Co-Principal Investigator |
| CRF | Case Report Form |
| d | days |
| DCA | dual-cure activator |
| DD | device deficiency |
| EC | Ethics Committee |
| eCRF | electronic Case Report Form |
| FDA | Food & Drug Administration |
| FDI | Fédération Dentaire Internationale (World Dental Federation) |
| GCP | good clinical practice |
| GI | glass ionomer |
| HIPAA | Health Insurance Portability and Accountability Act |
| ICF | informed consent form |
| IDE | investigational device exemption |
| IRB | Institutional Review Board |
| mos | months |
| MP | Monitoring Plan |
| PHI | Personal Health Information |
| SAP | Statistical Analysis Plan |
| SADE | serious adverse device effect |
| SAE | serious adverse event |
| SE | self-etch |
| SBU | Scotchbond <sup>TM</sup> Universal |
| SBU+ | Scotchbond <sup>TM</sup> Universal Plus |
| SOP | standard operating procedure |
| TE | total-etch |
| USADE | unanticipated serious adverse device effect |
| yr | year |

CLIN-PROT-CIP-11-050069


#### **TABLE OF CONTENTS**

| 1. | | PSIS | |
|---|---|---|---|
| 2. | IDEN | TIFICATION AND DESCRIPTION OF THE INVESTIGATIONAL DEVICE | .14 |
| 2.1 | | evice Regulatory Classification | 15 |
| 2.2 | 2 In | ntended Use of Device | 15 |
| 3. | JUST | IFICATION FOR THE STUDY DESIGN OF THE CLINICAL | |
| INVI | ESTIG | ATION | 16 |
| 3.1 | l B | ackground | 16 |
| 3.2 | 2 R | ationale For Studying The Specific Population/Condition | 18 |
| 3.3 | 3 R | ationale For Study Design | 18 |
| 4. | BENE | EFITS AND RISKS OF THE INVESTIGATIONAL DEVICE, CLINICAL | |
| PRO | CEDU | RE, AND CLINICAL INVESTIGATION | 19 |
| 4.] | l B | enefits of the Device | 19 |
| 4.2 | 2 R | isks of the Device | 19 |
| 4.3 | 3 A | nticipated Adverse Device Effects | 19 |
| 4.4 | 4 R | esidual Risks | 19 |
| 4.5 | 5 R | isk of Interactions with Concomitant Medical Treatments | 19 |
| 4.6 | 6 M | litigation of Risk | 20 |
| 4.7 | 7 R | ationale for Benefit-Risk Ratio | 20 |
| 5. | OBJE | CTIVES OF THE CLINICAL INVESTIGATION PLAN | 20 |
| 5.1 | l P | urpose | 20 |
| 5.2 | 2 P | rimary Objective | 20 |
| 5.3 | 3 E | ndpoints | 21 |
| | 5.3.1 | Primary Endpoints | 21 |
| | 5.3.2 | Secondary Endpoints | 21 |
| | 5.3.3 | Safety Endpoints | 21 |
| 6. | DESIG | GN OF CLINICAL INVESTIGATION | 22 |
| 6.1 | l D | esign | 22 |
| 6.2 | 2 In | nvestigational Device(s) and Comparator(s) | 22 |
| 6.3 | 3 S | ubject Enrollment | 23 |
| | 6.3.1 | Enrollment Criteria | 23 |
| 6.4 | 1 P | rocedures and Assessments | 25 |
| | 6.4.1 | Procedures and Assessments Diagram | 25 |
| | 6.4.2 | Informed Consent Process | 26 |
| | 6.4.3 | Demographics and Subject Characteristics | 26 |
| | 6.4.4 | Vital Signs | |
| | 6.4.5 | Randomization | 27 |
| | 6.4.6 | Intra-oral photographs | 27 |
| | 6.4.7 | Restoration and Application of Study Treatments | |

CLIN-PROT-CIP-11-050069

| 6.4.8 | Post-Restoration Assessments | 28 |
|---|---|---|
| 6.4.9 | Adverse Events and Adverse Device Effects | 34 |
| 6.4.10 | Prohibited Procedures and Treatments | 34 |
| 6.4.11 | End of Study Documentation | 34 |
| 6.5 S | ubject Withdrawal | 34 |
| 6.5.1 | Reasons for Subject Withdrawal | 34 |
| 6.5.2 | Reasons for Tooth Withdrawal | 35 |
| 6.5.3 | Handling of Withdrawal or Termination | 35 |
| 6.6 V | ISIT SCHEDULE AND DESCRIPTION OF STUDY VISITS | 36 |
| 6.6.1 | Point of Enrollment | 36 |
| 6.6.2 | Visits | 36 |
| 6.6.3 | Point of Exit | 39 |
| 6.7 R | ole of Sponsor Representation | 39 |
| 6.7.1 | Monitoring | 39 |
| 6.7.2 | Other Sponsor Oversight | 40 |
| 7. STAT | ISTICAL DESIGN AND ANALYSIS | 40 |
| 7.1 S | tatistical Hypotheses | 41 |
| 7.2 Sa | ample Size Determination | 41 |
| 7.3 P | opulation for Analyses | 41 |
| 7.4 S <sub>1</sub> | tatistical Analyses | 41 |
| 7.4.1 | Demographics and Baseline Characteristics | 42 |
| 7.4.2 | Analysis of Primary Endpoints | |
| 7.4.3 | Analysis of Secondary Endpoints | |
| 7.4.4 | Analysis of Safety Endpoint | 43 |
| 7.5 P | lanned Interim Analyses and Criteria for Clinical Investigation | 43 |
| 7.6 Pr | rocedures for Missing, Unused or Spurious Data | 43 |
| | rocedures for Reporting Deviations from Statistical Plan | 43 |
| | alidation Plan | 44 |
| 8. DATA | A MANAGEMENT | 44 |
| 8.1 D | ata Collection and Management Responsibilities | 44 |
| | tudy Records Retention | 44 |
| 8.3 S | ponsor Oversight | 45 |
| 9. AME | NDMENTS TO THE CIP | 45 |
| 10. DEVI | ATIONS FROM THE CIP | 45 |
| 10.1 D | reviation Reporting Timelines | 46 |
| 11. DEVI | CE ACCOUNTABILITY | 46 |
| 11.1 D | evice Labeling | 47 |
| | dditional Study-Specific Equipment/Device(s) | 48 |
| | EMENTS OF COMPLIANCE | 48 |

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069

| 12.1 | Ethical Considerations | 48 |
|---|---|---|
| 12.2 | Periodic Reviews | 48 |
| 12.3 | Participant Confidentiality | 48 |
| 12.4 | Conflict of Interest | 49 |
| 12.5 | Insurance | 49 |
| 13. AD | VERSE EVENTS, ADVERSE DEVICE EFFECTS, AND DEVICE | |
| DEFICIE | ENCIES | 50 |
| 13.1 | Safety and Event Reporting Definitions | 50 |
| 13.2 | Classification of Events | 51 |
| 13.2 | 2.1 Severity Ratings | 51 |
| 13.2 | 2.2 Relatedness to Study Treatment | 51 |
| 13.3 | Reporting Timelines | 52 |
| 13.4 | Details Concerning Safety Recording and Reporting Requirements | 53 |
| 13.4 | l.1 Investigator | 53 |
| 13.4 | I.2 Sponsor | 53 |
| 13.5 | Anticipated Adverse Events and Adverse Device Effects | 54 |
| 14. VU | LNERABLE POPULATION | 54 |
| 15. SU | SPENSION OR PREMATURE TERMINATION OF THE CLINICAL | |
| INVEST | IGATION PLAN | 55 |
| 15.1 | .1 By Sponsor | 56 |
| 15.1 | .2 By IRB | 56 |
| 16. RE | GISTRATION AND PUBLICATION POLICY | 56 |
| 16.1 | Public Registration | 56 |
| 16.2 | Publications Resulting From Study | 56 |
| | BLIOGRAPHY | 56 |
| 18. ST | UDY-SPECIFIC APPENDICES | 59 |
| 18.1 | Appendix A. American Association of Anesthesiologists (ASA) Physical Sta | tus |
| Classi | fication System | 60 |
| 18.2 | Appendix B. Grace and Smales Mobility Index | 61 |
| 18.3 | Appendix C. ICDAS Radiographic Scoring System | 62 |
| 18.4 | Appendix D. Revision History | 63 |

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


#### 1. SYNOPSIS

| Study Title | Prospective, randomized, split-mouth study evaluating the clinical performance of a new dental adhesive, $3M^{TM}$ Scotchbond <sup>TM</sup> Universal Plus Adhesive, compared to $3M^{TM}$ Scotchbond <sup>TM</sup> Universal Adhesive when used for posterior Class I and Class II restorations with $3M^{TM}$ Filtek <sup>TM</sup> Universal Restorative |
|---|---|
| Study Type | Post-market, interventional |
| Principal<br>Investigator (PI) | Name: Jorge Perdigao, DMD, MS, PhD Title: Professor Site: University of Minnesota |
| Co-Principal<br>Investigator<br>(Co-PI) | Name: Hooi Pin Chew (BDS, FDSRCS, PhD) Title: Associate Professor Site: University of Minnesota |
| Co-Investigators | Name: Erin C. Westmeyer (DDS) Title: Clinical Assistant Professor Site: University of Minnesota |

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069

| | Names Ignative V. Lee (DDC MC) |
|---|---|
| | Name: Ignatius K. Lee (DDS, MS) Title: Clinical Associate Professor |
| | Site: University of Minnesota |
| | Department of Restorative Sciences |
| | Office Address: |
| | 16-256B Moos Tower |
| | 515 Delaware St. SE |
| | Minneapolis, MN 55455 |
| | Email: |
| | Telephone: |
| | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| | Name: Brian Hatch (DDS) |
| | Title: Clinical Assistant Professor |
| | Site: University of Minnesota |
| | Department of Primary Dental Care |
| | Office Address: |
| | 9-268 Moos Tower |
| | 515 Delaware St. SE |
| | Minneapolis, MN 55455 |
| | Email: |
| | Telephone: |
| Device under<br>Investigation<br>Summary | The investigational device in this study is Scotchbond <sup>TM</sup> Universal Plus (SBU+) Adhesive, which is manufactured by 3M. It is a light-curing, single-component dental adhesive that is compatible with light-, dual-, and self-cure composite filling materials, cements, and core build-up materials. The adhesive can be used for "self-etch" procedures, selective enamel etching procedures, or "total-etch/etch-and-rinse" procedures, and a separate dual-cure activator (DCA) is not necessary. The intended purpose of SBU+ Adhesive is to be used as a bond-promoting substance between the tooth and dental restorations. It may also be used as a dentin sealant and as a bonding agent for repair of restorations. The intended users of Scotchbond <sup>TM</sup> Universal Plus Adhesive are qualified dental professionals who have theoretical and practical knowledge on usage of dental products. |
| Sponsor | 3M<br>3M Healthcare Business Group<br>3M Center – 270-4N<br>St. Paul, MN. 55144 |
| Purpose | The purpose of this study is to confirm the clinical effectiveness of Scotchbond <sup>TM</sup> Universal Plus Adhesive by comparing it with the predicate adhesive device. |

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069

| Design | This is a prospective, randomized, controlled, open-label, assessorblinded, split-mouth, single-center post-market clinical follow-up study. The study will enroll a minimum of 50 Subjects. |
|---|---|
| Selection of<br>Subjects | To be considered eligible for randomization, Subjects must meet all the inclusion criteria and none of the exclusion criteria. Subjects are to be assessed for eligibility no more than 21 days prior to the planned oral care procedures, and eligibility will be confirmed on the day of the restorations. If, for any reason, a Subject's restorative appointment is delayed beyond 21 days after consent, then the Subject will be reassessed to ensure that they still meet the eligibility criteria. Subjects who have provided informed consent but who do not meet all eligibility criteria at the time of the restorations will not be eligible for randomization, will not qualify for participation in the study, and will be considered a screening failure. |
| | <ol> <li>Inclusion Criteria:</li> <li>Inclusion criteria include the following: <ol> <li>The Subject is between the ages of 18 and 70 years old at time of consent.</li> <li>The Subject requires at least two direct composite restorations for posterior Class I or Class II carious lesions in vital teeth that are asymptomatic and with minimal mobility (&lt; 1 mm in the buccolingual direction).</li> <li>Study teeth have a minimum buccolingual diameter of the occlusal surface that is at least 1/3 of the distance between the buccal and lingual cusps.</li> </ol> </li> <li>Teeth selected for Class II restorations need to have an adjacent tooth in a position that will allow for a contact relationship to be established.</li> <li>The Subject is able and willing to sign Informed Consent Form in English without assistance.</li> <li>The Subject is able and willing to be available for all scheduled study visits.</li> <li>The Subject is in good general health (ie, meets ASA Level I or ASA Level II classification criteria).</li> <li>The selected teeth need to have occlusal contact with an antagonistic natural tooth.</li> <li>The Subject has existing radiographic images of the study teeth of current and acceptable diagnostic quality obtained within the previous 12 months.</li> </ol> |

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069

| | Exclusion Criteria: |
|---|---|
| | Preoperative exclusion criteria include the following: |
| | 1. The Subject has a history of adverse reaction to any materials |
| | used in this study. |
| | 2. The Subject is pregnant or breast feeding at the time of screening. |
| | 3. The Subject has fewer than 20 teeth. |
| | 4. The Subject is taking part in or planned to be enrolled in an |
| | evaluation of other restorative materials at any time during |
| | the study. |
| | <ol> <li>The Subject has advanced periodontal disease (ie, Grace &amp;<br/>Smales Mobility Index grade ≥ 2) that involve the study</li> </ol> |
| | teeth. |
| | 6. The Subject had orthodontic appliance treatment within the previous 3 months. |
| | 7. The Subject has pronounced enamel wear facets, indicting |
| | severe, on-going bruxism. 8. The Subject has severe xerostomia. |
| | 9. The study tooth has a history of or existing, prolonged tooth |
| | hypersensitivity. |
| | 10. The study tooth is an abutment for fixed or removable |
| | prostheses. |
| | 11. The study tooth has a fracture or is visibly cracked such that it may impact the longevity of the tooth. |
| | 12. The carious lesion is stage RC5 or RC6 of the ICDAS |
| | radiographic scoring system. |
| | 13. The Subject is unable to understand study procedures or |
| | provide consent in English. |
| | 14. The Subject is an employee or student of the study investigator(s). |
| | Intraoperative exclusion criteria include the following: |
| | The Subject has pulp exposure of either study tooth during |
| | restoration procedure. |
| | In accordance with regulation number 21CFR872.3200 from the |
| | United States Food & Drug Administration (FDA), Scotchbond™ |
| | Universal Plus Adhesive is a 510(k)-cleared, Class II device |
| Device Regulatory | (K192961) with the following indication for use: |
| Classification | |
| | Direct Indications: |
| | Bonding for all methacrylate-based light-, dual-, and self-cure Bonding for all methacrylate-based light-, dual-, and self-cure |
| | composite or compomer filling materials |

| <b>3M</b> |
|------------|
| HealthCare |

CLIN-PROT-CIP-11-050069

| | 7 2 4 |
|---|---|
| | Root surface desensitization |
| | Bonding of methacrylate-based fissure sealants |
| | Protective varnish for glass ionomer fillings |
| | Repair of composite and compomer fillings |
| | Sealing of cavities prior to placement of amalgam restorations |
| | Indirect Indications: |
| | <ul> <li>Cementation of indirect restorations in combination with<br/>RelyX Universal and other resin cements (follow applicable<br/>Instructions for Use)</li> </ul> |
| | <ul> <li>Bonding for all methacrylate-based light-, self-, and dual-cure<br/>core build-up materials and cements</li> </ul> |
| | Cementation of veneers when combined with RelyX Veneer<br>Cement |
| | <ul> <li>Intraoral repair of composite restorations, porcelain fused to metal, and all-ceramic restorations without extra primer</li> <li>Sealing of cavities and preparation of tooth stumps prior to temporary cementation of indirect restorations</li> </ul> |
| Primary<br>Objective(s) | The primary objective of this study is to compare the clinical efficacy of Scotchbond <sup>TM</sup> Universal Plus Adhesive with Scotchbond <sup>TM</sup> Universal Adhesive when used in self-etch mode for preparation of posterior Class I and Class II restorations using Filtek <sup>TM</sup> Universal Restorative material in adult patients. |
| | Primary Endpoint: |
| | The primary endpoints, which are based partly on the FDI World Dental Federation criteria, are the following criteria at the final assessment (24 months): |
| | <ul> <li>the proportion of Subjects with partial or complete loss of the restoration materials</li> <li>fracture grade</li> </ul> |
| <b>-</b> • • · · · · | marginal adaptation grade |
| Endpoint(s) | Secondary Endpoints: |
| | The secondary endpoints are the following modified FDI World Dental Federation criteria: |
| | • the proportion of Subjects with partial or complete loss of the restoration materials at 6 months and 12 months |
| | <ul> <li>time to restoration failure (ie, time to partial or complete loss of restoration)</li> <li>fracture grade at 6 months and 12 months</li> </ul> |
| | - Tractare grade at 6 months and 12 months |



CLIN-PROT-CIP-11-050069

| | <ul> <li>marginal adaptation grade at baseline, 6 months, and 12 months</li> <li>approximal anatomical form (contact point) grade at baseline, 6 months, 12 months, and 24 months</li> <li>incidence of recurrent caries at 6 months, 12 months, and 24 months</li> <li>marginal staining grade at baseline, 6 months, 12 months, and 24 months</li> <li>surface staining grade at baseline, 6 months, 12 months, and 24 months</li> <li>color match and translucency grade at baseline, 6 months, 12 months, and 24 months</li> <li>surface luster grade at baseline, 6 months, 12 months, and 24 months</li> <li>postoperative hypersensitivity and tooth vitality grade at 6 months, 12 months, and 24 months</li> </ul> |
|---|---|
| | Safety Endpoints: The safety endpoint is the incidence of Adverse events (AEs). |
| | Subjects who satisfy all inclusion criteria and none of the exclusion criteria and who have provided informed consent will be eligible for randomization, which will occur immediately after teeth preparation but before the initial application of any adhesive agent. A unique Subject identification number will be assigned upon enrollment, and study data will be reported according to this unique Subject identifier. The unique Subject identification number will not contain information that could identify the Subject. |
| Randomization | Randomization of the premolars or molars, which will be numbered using the Universal Numbering System (premolars = 4-5, 12-13, 20-21, or 28-29; molars = 1-3, 14-16, 17-19, or 30-32), to study treatments will be centralized and electronic. Either two pre-molars or two molars from each Subject will be randomized in a 1:1 ratio such that one of the teeth will be randomized to undergo restoration using SBU+ Adhesive (Treatment), and the other tooth will undergo restoration using SBU Adhesive (Control). Study teeth will be assigned randomization numbers starting with the lowest tooth number. The first material for assignment according to the randomization schedule will be assigned to the lower tooth number in the pair. |

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


| | The entire duration of the study is expected to last approximately 3 years, with individual Subject participation expected to last up to 2 years ( $\pm$ 45 days). |
|---|---|
| Duration of the Study | <ul> <li>Subject participation will include the following:</li> <li>Screening visit (no more than 21 days before tooth restoration)</li> <li>Restoration procedures and baseline assessments – Day 0</li> <li>Follow-up visits after the restorations at: <ul> <li>6 months (± 14 days)</li> <li>1 year (± 30 days)</li> <li>2 years (± 45 days)</li> </ul> </li> </ul> |
| | Subjects may participate in additional unscheduled visits as required during the study if evaluation of any study tooth is required outside of the scheduled study visits. |
| Sponsor Study<br>Contact | Name: Paula Myhre (Clinical Project Manager and Study Monitor) Address: 3M Center, 270-4N-04 St. Paul, MN 55144-1000 Telephone: Email: |
| Medical Monitor<br>Contact | Name: Dr. Andreas Syrek Address: 3M Deutschland GmbH, ESPE Platz 82229 Seefeld, Germany Telephone: Email: |

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 

## CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


## 2. IDENTIFICATION AND DESCRIPTION OF THE INVESTIGATIONAL DEVICE

The investigational device in this study is Scotchbond™ Universal Plus (SBU+) Adhesive, which is manufactured by 3M (Table 2-1). SBU+ Adhesive is a light-curing, single-component dental adhesive that is compatible with light-, dual-, and self-cure composite filling materials, cements, and core build-up materials. The adhesive can be used for "self-etch" procedures, selective enamel etching procedures, or "total-etch/etch-and-rinse" procedures, and a separate dual-cure activator (DCA) is not necessary. SBU+ Adhesive is radiopaque (radiopacity similar to dentin) and the formulation is bisphenol-A (BPA)-derivative free. The intended purpose of SBU+ Adhesive is to be used as a bond-promoting substance between the tooth and dental restorations. It may also be used as a dentin sealant and as a bonding agent for repair of restorations. The intended users of SBU+ Adhesive are qualified dental professionals who have theoretical and practical knowledge on usage of dental products.

The comparator product (ie, Control product) for the investigational device will be Scotchbond<sup>TM</sup> Universal (SBU) Adhesive, which is also manufactured by 3M (Table 2-1). SBU Adhesive bonds methacrylate-based restoratives, cement and sealant materials to dentin, enamel, glass ionomer and various indirect restorative substrates (metals, glass ceramics, alumina, and zirconia) without an extra primer step. SBU Adhesive can be used reliably in totaletch, self-etch or selective-etch mode for both direct and indirect restorations. The primary use is with light-cured materials, however, when used in conjunction with a separate activation solution, Scotchbond<sup>TM</sup> Universal DCA Dual Cure Activator, it has the capability to also bond to self- or dual-cure composite and cement materials that rely on self-cure polymerization. In this study, the comparator product will be applied and polymerized using a curing light before applying 3M<sup>TM</sup> Filtek<sup>TM</sup> Universal Restorative.

**Table 2-1: Device Information** 

| Investigational | Device | Comparator Device | |
|---|---|---|---|
| Device Name | Manufacturer | Device Name | Manufacturer |
| Scotchbond™ Universal<br>Plus Adhesive | 3M | Scotchbond™<br>Universal Adhesive | 3M |

## CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


#### 2.1 DEVICE REGULATORY CLASSIFICATION

In accordance with regulation number 21CFR872.3200 from the United States Food & Drug Administration (FDA), SBU+ Adhesive is a 510(k)–cleared, Class II device (K192961) with the following indication for use:

#### **Direct Indications**:

- Bonding for all methacrylate-based light-, dual-, and self-cure composite or compomer filling materials
- Root surface desensitization
- Bonding of methacrylate-based fissure sealants
- Protective varnish for glass ionomer fillings
- Repair of composite and compomer fillings
- Sealing of cavities prior to placement of amalgam restorations

#### **Indirect Indications:**

- Cementation of indirect restorations in combination with RelyX Universal and other resin cements (follow applicable Instructions for Use)
- Bonding for all methacrylate-based light-, self-, and dual-cure core build-up materials and cements
- Cementation of veneers when combined with RelyX Veneer Cement
- Intraoral repair of composite restorations, porcelain fused to metal, and allceramic restorations without extra primer
- Sealing of cavities and preparation of tooth stumps prior to temporary cementation of indirect restorations

#### 2.2 INTENDED USE OF DEVICE

For the teeth of Subjects in this study that are randomized into the Treatment arm, SBU+ Adhesive will be applied and polymerized using a curing light before applying 3M<sup>™</sup> Filtek<sup>™</sup> Universal Restorative. For this study, SBU+ Adhesive will be used in accordance with its cleared labeling and indications for use and is, therefore, exempt from the investigational device exemptions (IDE) regulation because it meets the conditions for an exempt investigation as provided in paragraph C of 21CFR812.2 from the FDA. The indications, precautionary measures, and instructions can be found in the IFU document for SBU+ Adhesive (3M).

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


## 3. JUSTIFICATION FOR THE STUDY DESIGN OF THE CLINICAL INVESTIGATION

#### 3.1 BACKGROUND

#### Class I and Class II Dental Caries

Class I and Class II dental caries lesions occur on various surfaces of the mandibular and maxillary posterior teeth (ie, premolars and molars) and can range in severity from incipient to severe. Direct restoration of posterior tooth caries, which is the focus of this study, have traditionally involved the use of amalgam fillings. However, the use of resin composites, which are chemically and micromechanically bound to the dentin and enamel by dental resin adhesives<sup>2</sup>, to restore posterior tooth caries has increased over the past few decades due in part to the poor esthetics of amalgam and concerns about mercury content in amalgam alloys. Since dental resin adhesives are known to critically impact the performance of resin restorations<sup>2</sup>, this study focuses on retention, fracture, and marginal integrity (ie, marginal adaptation) when using two different dental resin adhesives to bond a resin composite to the dentin and enamel of Class I and Class II carious lesions.

#### Resin Composite Restorations on Posterior Teeth

Resin composite restorations, like all restorations, undergo extreme challenges in the oral cavity, including mechanical degradation (eg, thermocycling from hot and cold food and beverage consumption), chemical and biochemical degradation, short-term elution of unreacted composite monomers, and long-term enzymatic breakdown due, in part, to hydrolase/esterase activity in the oral cavity.<sup>2</sup> For these reasons and others, composite restoration failure is a major concern and can lead to costly repair or replacement of the restoration, potentially more costly treatments (eg, root canal therapy), or eventual loss of the tooth.<sup>2</sup>

A 2015 meta-analysis of posterior teeth restorations using either amalgam or composite resin, showed a mean annual fail rate (AFR) for composite resin restorations of 3.17%.<sup>3</sup> A meta-analysis of longitudinal studies with at least a 5-year follow-up for composite restorations of posterior teeth showed an AFR of 1.8% for all restorations analyzed and a 3.2%-3.5% AFR for medium-caries-risk to high-caries-risk patients.<sup>4</sup> Similarly, two single-center studies of restorations for Class II caries reported an AFR of composite restorations ranging from 1.78% to 2.9%.<sup>5, 6</sup> The leading cause for restoration failure in posterior teeth was secondary caries occurring at the margin between the restoration materials and the remaining tooth.<sup>5</sup>

#### Classification of Dental Resin Adhesives & Retention in Class I and Class II Restorations

Contemporary dental resin adhesives are generally classified by their mode of application, including the following: (i) self-etch (SE) adhesives, which use a non-rinse acidic monomer to

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 



CLIN-PROT-CIP-11-050069


simultaneously condition and prime the enamel/dentin; (ii) total etch (TE) adhesives, also known as etch-and-rinse adhesives, which involved the application of phosphoric acid followed by rinsing; (iii) selective etch adhesives, whereby an etch/rinse application occurs only on the enamel surrounding a lesion; and (iv) glass ionomer (GI) adhesives, which micromechanically bond to the tooth structure following a mild acid pre-treatment.<sup>2, 7</sup>

To date, there have been several publications describing comparative prospective studies or randomized controlled trials focused on comparing different types of contemporary adhesives (eg, SE vs TE vs GI) when used for posterior tooth restorations. 8-13 Four of these studies 8, 10, 11, 13 used USPHS scoring criteria (ie, Alfa, Beta, or Charlie, with Alfa being "Excellent" to compare restorations using different types of contemporary adhesives, and one study<sup>12</sup> used FDI scoring criteria (ie, ranging from 1-5 with a score of 1 being "Excellent" and 5 being "Poor"<sup>15</sup>) to compare restorations. One study used both USPHS and FDI criteria to score restorations. 9 Of these 6 publications, only 2 assessed functionality of the restorations placed using different adhesives related to retention, fracture, and marginal adaptation (ie, marginal integrity) after 2 years; 8, 10 the others assessed functionality (ie, retention, fracture, or marginal adaptation) after 1 year 11-13 or after 1 year to 20 months9. Using USPHS scoring criteria, retention scores of Alfa for restorations using two different TE adhesives (3M<sup>TM</sup> Adper<sup>TM</sup> Scotchbond<sup>TM</sup> 1 XT and Bisco One-Step<sup>TM</sup> Plus) were 100% after 2 years, while retention scores of Alfa for restorations using 4 different types of SE adhesives (3M<sup>TM</sup> Adper<sup>TM</sup> Scotchbond<sup>TM</sup> SE, 3M<sup>TM</sup> Adper<sup>TM</sup> Prompt<sup>TM</sup> L-Pop, Kuraray CLEARFIL<sup>TM</sup> S<sup>3TM</sup> Bond, or Heraeus Kulzer iBond<sup>TM</sup>) ranged from 90.5% to 92%.<sup>8, 10</sup> In these two studies, marginal adaptation scores of Alfa after 2 years were reported to range from 9.5% to 66.7% for restorations using the 4 different types of SE adhesives, whereas restorations placed with the two different TE adhesives ranged from 83.3% to 87%. 8, 10 In one of the studies, Perdigao et al, the percentage of restorations with a fracture score of Alfa after 2 years was similarly lower (90.5% to 92%) when the restoration included the SE adhesives vs when the restoration included the TE adhesive (100%).<sup>10</sup>

#### Scotchbond™ Universal Adhesives

Scotchbond™ Universal Plus (SBU+) Adhesive, which is based on the chemistry of a predicate device, Scotchbond™ Universal (SBU) Adhesive, is a multimode dental resin adhesive that can be used in self-etching or total-etching (with or without selective enamel etching) procedures. While there have been no publications regarding clinical studies of SBU+ Adhesive, there has been 1 publication reporting on the laboratory evaluation of SBU Adhesive on extracted human teeth (ie, *ex vivo* study) and 16 publications reporting on clinical trials that included the use of SBU Adhesive. 9, 13, 16-29 The *ex vivo* study assessed microtensile bond strength, nanoleakage, and *in situ* degree of conversion using extracted, caries-free, human third molars. 22 Two



CLIN-PROT-CIP-11-050069


publications were related to the treatment of caries in primary teeth, with one of the publications being a trial design only<sup>19, 23</sup>, and 11 publications reported the use of SBU Adhesive in restoration of NCCLs. <sup>16-18, 20, 21, 24-29</sup> The remaining two publications reported on Class I and Class II cavity restorations. <sup>9, 13</sup>

Balkaya et al compared a micro-hybrid composite resin with a bulk-fill composite resin and high-viscosity GI cement when used to restore Class II restorations; in this study, SBU Adhesive was used for both a micro-hybrid composite resin and a bulk-fill composite resin, but there was no mention of whether SBU Adhesive was applied using an SE or a TE procedure. In contrast, Carvalho et al compared Class I and Class II restorations using SBU Adhesive applied via total etching (TE), via self-etching (SE), or via selective enamel etching. After 12 to 20 months, 100% of the restorations were scored as acceptable, having a USPHS score of Alfa, for retention. In addition, 45 of 46 (97.8%) restorations using SBU Adhesive via SE had a fracture score of Alfa after 12 to 20 months, and the 92 teeth that had been restored using SBU Adhesive applied via TE (n = 46) or using SBU Adhesive applied via selective enamel etching (n = 46) had fracture scores of Alfa (100%). Marginal adaptation scores after 12-20 months for teeth that had been restored using SBU Adhesive were: TE = 45 of 46 with score of Alfa (97.8%); SE = 44 of 46 with a score of Alfa (95.7%); and Selective enamel etching = 45 of 46 with a score of Alfa (97.8%).

#### 3.2 RATIONALE FOR STUDYING THE SPECIFIC POPULATION/CONDITION

Subjects with Class I or Class II carious lesions (ie, in molars or premolars) were selected as the specific population/condition for this study since these types of caries have been reported to account for 68.5% of all dental caries<sup>30</sup>, making restorations for posterior teeth caries a frequently performed procedure for dental practitioners.

#### 3.3 RATIONALE FOR STUDY DESIGN

To have a high level of evidence, a prospective, controlled, within-subject, randomized, single center trial was the design selected for this study. The within-subject design includes randomizing one tooth of a Subject to the Treatment arm and one other tooth to the Control arm, thereby allowing each Subject to be exposed to both treatment arms. SBU Adhesive was selected as the comparator (Control product) as it is the predicate device for SBU+ Adhesive and, as mentioned in Section 3.1, has been studied previously in self-etch and total-etch mode restorations of Class I and Class II restorations. SE mode restorations have been selected for this study based on a previous study showing that Class I/Class II restorations using SBU Adhesive applied via SE mode or applied via TE mode have similar retention rates, and SE mode does not require the use of an additional variable (an acid etchant). To further limit study variables, Filtek Universal Restorative material will be used for both the Treatment arm and



CLIN-PROT-CIP-11-050069


the Control arm, which will allow for the collection of information related to this composite resin.

The primary endpoints of this study are restoration retention, fracture, and marginal adaptation scoring since the purpose of this study is to compare SBU+ Adhesive with its predicate device (SBU Adhesive) in relation to functional aspects of the restorations. The follow-up period of 24 months was selected based on previous 2-year studies of other composite resin adhesives showing differences in retention, fracture, and marginal adaptation scoring.<sup>8, 10</sup>

## 4. BENEFITS AND RISKS OF THE INVESTIGATIONAL DEVICE, CLINICAL PROCEDURE, AND CLINICAL INVESTIGATION

#### 4.1 BENEFITS OF THE DEVICE

The clinical benefit of the investigational device (SBU+ Adhesive) and the control device (SBU Adhesive) is that they hold direct restorations in place, hold indirect restorations in place when used in combination with a luting agent, and help in sealing and desensitization.

#### 4.2 RISKS OF THE DEVICE

Dental adhesives are commonly used medical devices throughout dental care settings that have resulted in few problems. A potential risk to the Subjects in this study includes an allergic reaction by skin contact. If an allergic reaction occurs, the Subject should seek medical attention as needed, the product should be removed if necessary, and future use of the device should not occur.

#### 4.3 ANTICIPATED ADVERSE DEVICE EFFECTS

Due to substances in the investigative device and the comparator device used for this study, it is anticipated that the device may cause an allergic reaction by skin contact in certain individuals. Symptoms of allergic reactions (eg, erythema) are being captured as adverse events in this study.

#### 4.4 RESIDUAL RISKS

The Subjects will undergo long-term exposure to polymerized material, including polymerized acrylate, which is more inert (ie, less sensitizing) than monomeric acrylate. Therefore, residual risks are expected to be minimal.

#### 4.5 RISK OF INTERACTIONS WITH CONCOMITANT MEDICAL TREATMENTS

There is minimal risk of interaction between the investigative device or the comparator device and concomitant medical treatments. The manufacturer advises against the use of substances

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 



CLIN-PROT-CIP-11-050069


such as desensitizers, disinfectants other than chlorhexidine-containing agents, astringents, dentin sealants, and rinsing solutions before applying SBU+ Adhesive as residues of these substances can be detrimental to the bonding strength of the device. Only chlorhexidine-containing solutions are permitted during cavity/tooth preparation prior to restoration in this study (see Section 6.4.7.1).

#### 4.6 MITIGATION OF RISK

Risk related to the device may be mitigated or controlled through appropriate selection of study Subjects for inclusion into this study, adherence to this Clinical Investigation Plan (CIP), and reporting of Adverse Events (AEs), Device Deficiencies (DDs), and deviations to the Sponsor. For example, Subjects with known acrylate allergies are excluded from participating in this study (see Section 0).

#### 4.7 RATIONALE FOR BENEFIT-RISK RATIO

Insertion of direct restorations is a standard of care in dentistry. All products used in this study are commercially available, have regulatory clearance (e.g. 510K, CE mark), will be used per their respective Instructions for Use including the indications, and thus can be used for routine clinical treatment.

Based upon the risks and benefits listed above and adherence to this CIP, the study Subjects are at no greater risk of harm than individuals being treated for similar lesions who are not participating in this study. The use of SBU+ Adhesive is being used in accordance with its intended use consistent with standard dental treatment plans for patients not participating in this study.

#### 5. OBJECTIVES OF THE CLINICAL INVESTIGATION PLAN

#### 5.1 PURPOSE

The purpose of this study is to confirm the clinical effectiveness of Scotchbond<sup>TM</sup> Universal Plus Adhesive by comparing it with the predicate adhesive device.

#### 5.2 PRIMARY OBJECTIVE

The primary objective of this study is to compare the clinical efficacy of Scotchbond<sup>TM</sup> Universal Plus Adhesive against Scotchbond<sup>TM</sup> Universal Adhesive when used in self-etch mode for preparation of posterior Class I and Class II restorations using Filtek<sup>TM</sup> Universal Restorative material in adult patients.

## CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


#### 5.3 ENDPOINTS

#### 5.3.1 Primary Endpoints

The primary endpoints, which are based partly on the FDI World Dental Federation criteria<sup>15</sup>, are the following criteria at the final assessment (24 months):

- the proportion of Subjects with partial or complete loss of the restoration materials
- fracture grade
- marginal adaptation grade

#### **5.3.2 Secondary Endpoints**

The secondary endpoints are the following modified FDI World Dental Federation criteria:

- the proportion of Subjects with partial or complete loss of the restoration materials at 6 months and 12 months
- time to restoration failure (ie, time to partial or complete loss of restoration)
- fracture grade at 6 months and 12 months
- marginal adaptation grade at baseline, 6 months, and 12 months
- approximal anatomical form (contact point) grade at baseline, 6 months, 12 months, and 24 months
- incidence of recurrent caries at 6 months, 12 months, and 24 months
- marginal staining grade at baseline, 6 months, 12 months, and 24 months
- surface staining grade at baseline, 6 months, 12 months, and 24 months
- color match and translucency grade at baseline, 6 months, 12 months, and 24 months
- surface luster grade at baseline, 6 months, 12 months, and 24 months
- postoperative hypersensitivity and tooth vitality grade at 6 months, 12 months, and 24 months

#### **5.3.3** Safety Endpoints

The safety endpoint is the incidence of AEs.

## CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


#### 6. DESIGN OF CLINICAL INVESTIGATION

#### 6.1 DESIGN

This is a prospective, randomized, controlled, open-label, assessor-blinded, split-mouth, single-center post-market clinical follow-up study. The study will enroll a minimum of 50 Subjects from a single site located in Minneapolis, Minnesota, USA. Each Subject will undergo restorations on two independent teeth (ie, two restorations) with each tooth restoration using only one type of adhesive. All teeth needing treatment that are not included in the study will be treated by the dentist using their standard of care.

Subjects will be seen during Screening (no more than 21 days before the restoration procedure), on the day of the restoration procedure (Day 0, baseline), 6 months ( $\pm$  14 days) after the restorations, 1 year ( $\pm$  30 days) after restorations, and 2 years after restorations ( $\pm$  45 days). Subjects may participate in additional unscheduled visits as required during the study if evaluation of any study tooth is required outside of the scheduled study visits. Unscheduled visits may be initiated by either the Investigator or the Subject. The entire duration of the study is expected to last approximately 3 years, with individual Subject participation expected to last up to 2 years ( $\pm$  45 days).

To help minimize or avoid bias in the study, randomization of study teeth will occur after teeth preparation (see Section 6.4.5) but before the initial application of any adhesive. All assessments will be performed by two dental examiners that are independent of the dentist that placed the restorations and are blinded to the treatment arms. All examiners will be trained and calibrated for the scoring criteria before any Subject assessment occurs (see Section 6.4.8 for descriptions of assessments), and examiners will be retrained and recalibrated if any new evaluator is added to the list of assessors. After the second examiner has completed their assessments, then the examiners will compare their evaluations and a consensus will be reached for each of the scoring criteria at each visit. A consensus will be reached before the Subject leaves the visit, and the consensus assessments will be entered into the Case Report Form (CRF).

#### 6.2 INVESTIGATIONAL DEVICE(S) AND COMPARATOR(S)

Restorations will include the use of 3M<sup>™</sup> Filtek<sup>™</sup> Universal Restorative to match and blend to the color of the surrounding dentition. On one tooth, the restorative material will be bonded with SBU+ Adhesive (Treatment arm), and restorative material on the other tooth will be bonded using SBU Adhesive (Control arm). Both adhesives will be applied using the self-etch mode.

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


#### 6.3 SUBJECT ENROLLMENT

Subject enrollment will remain open until a minimum of 50 subjects are enrolled and confirmed eligible (see Section 6.3.1).

#### 6.3.1 Enrollment Criteria

In order to be considered eligible for randomization, Subjects must meet all the inclusion criteria listed in Section 6.3.1.1 and none of the exclusion criteria listed in Section 0. Subjects should be assessed for eligibility no more than 21 days prior to the planned oral care procedures, and eligibility will be confirmed on the day of the restorations. If, for any reason, a Subject's restorative appointment is delayed beyond 21 days after consent, then the Subject will be reassessed to ensure that they still meet the eligibility criteria. Subjects who have provided informed consent but who do not meet all eligibility criteria at the time of the restorations will not be eligible for randomization, will not qualify for participation in the study, and will be considered a screening failure.

#### 6.3.1.1 INCLUSION CRITERIA

Subjects may be included that meet the inclusion criteria in Table 6.3.1.1-1.

Table 6.3.1.1-1: Inclusion Criteria

| Number | Inclusion Criteria |
|---|---|
| 1 | The Subject is between the ages of 18 and 70 years old at time of consent. |
| 2 | The Subject requires at least two direct composite restorations for posterior Class I or Class II carious lesions in vital teeth that are asymptomatic and with minimal mobility (< 1 mm in the buccolingual direction). |
| 3 | Study teeth have a minimum buccolingual diameter of the occlusal surface that is at least 1/3 of the distance between the buccal and lingual cusps |
| 4 | Teeth selected for Class II restorations need to have an adjacent tooth in a position that will allow for a contact relationship to be established. |
| 5 | The Subject is able and willing to sign Informed Consent Form in English without assistance. |
| 6 | The Subject is able and willing to be available for all scheduled study visits. |
| 7 | The Subject is in good general health (ie, meets ASA Level I or ASA Level II classification criteria) Section 18, Appendix A. |
| 8 | The selected teeth need to have occlusal contact with an antagonistic natural tooth. |

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 



CLIN-PROT-CIP-11-050069


| Number | Inclusion Criteria |
|---|---|
| 9 | The Subject has existing radiographic images of the study teeth of current and |
| | acceptable diagnostic quality obtained within the previous 12 months. |

#### 6.3.1.2 EXCLUSION CRITERIA

Subjects must be excluded from participating in this study if they meet any of the preoperative or intraoperative criteria listed in Tables 6.3.1.2-1 and 6.3.1.2-2.

Table 6.3.1.2-1: Preoperative Exclusion Criteria

| Number | Exclusion Criteria |
|---|---|
| 1 | The Subject has a history of adverse reaction to any materials used in this study. |
| 2 | The Subject is pregnant or breast feeding at the time of screening. |
| 3 | The Subject has fewer than 20 teeth. |
| 4 | The Subject is taking part in or planned to be enrolled in an evaluation of other restorative materials at any time during the study. |
| 5 | The Subject has advanced periodontal disease (ie, Grace & Smales Mobility Index grade $\geq$ 2) that involve the study teeth. Appendix B |
| 6 | The Subject had orthodontic appliance treatment within the previous 3 months. |
| 7 | The Subject has pronounced enamel wear facets, indicating severe, on-going bruxism. |
| 8 | The Subject has severe xerostomia. |
| 9 | The study tooth has a history of or existing, prolonged tooth hypersensitivity. |
| 10 | The study tooth is an abutment for fixed or removable prostheses. |
| 11 | The study tooth has a fracture or is visibly cracked such that it may impact the longevity of the tooth. |
| 12 | The carious lesion is stage RC5 or RC6 of the ICDAS radiographic scoring system. Section 18, Appendix C |
| 13 | The Subject is unable to understand study procedures or provide consent in English. |
| 14 | The Subject is an employee or student of the study investigator(s). |



CLIN-PROT-CIP-11-050069


Table 6.3.1.2-2: Intraoperative Exclusion Criteria

| Number | Exclusion Criteria |
|---|---|
| 1 | The Subject has pulp exposure of either study tooth during the restoration procedure. |

#### 6.4 PROCEDURES AND ASSESSMENTS

The following sections describe the study procedures and data that will be collected at each visit for the duration of the study. The data listed below, and any relevant safety data will be collected during this study.

#### 6.4.1 Procedures and Assessments Diagram



# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


#### **6.4.2** Informed Consent Process

Informed Consent must be obtained for each Subject that meets eligibility criteria prior to any study activities being performed or data being collected. The Investigator or designee will review all relevant aspects of the study with the potential Study subject that are relevant to the Subject's decision to participate throughout the study. The Investigator or designee will provide ample time for the Subject to read and understand the IRB-approved ICF and to consider participation in the study.

The study Subject and the Investigator (or qualified designee) must sign and date the ICF. The Investigator or designee must file the original ICF and provide the Subject with a copy of the signed and dated ICF and any other written documentation per IRB/EC requirements. Subject privacy language (ie, HIPAA) per local regulations may be added to the local ICF by the Investigator.

The Informed Consent Process must be documented by the Investigator or designee. The Informed Consent Process includes documentation of the discussion regarding study procedures, Subject concerns, that the Subject was provided ample time to consider participation, and that all questions were answered prior to participation in any research activity.

In order to minimize pressure and undue influence on vulnerable Subjects (see Section 14), the Investigator or designee who is obtaining Informed Consent should ensure appropriate communication technique, such as avoidance of jargon and using plain language.

#### 6.4.3 Demographics and Subject Characteristics

After a Subject signs the informed consent form (ICF; see Section 6.4.2) and before the initial tooth restoration, the following demographic data and Subject characteristics will be collected and documented:

- Age
- Sex
- Race
- Ethnicity
- Tooth numbers for treated teeth
- Date of restoration

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


#### 6.4.4 Vital Signs

No vital signs (eg, height/weight) or laboratory assessments will be captured as part of this study.

#### 6.4.5 Randomization

Subjects who satisfy all inclusion criteria and none of the exclusion criteria and who have provided informed consent will be eligible for randomization, which will occur immediately after teeth preparation (see Section 6.4.7) but before the initial application of any adhesive agent. A unique Subject identification number will be assigned upon enrollment, and study data will be reported according to this unique Subject identifier. The unique Subject identification number will not contain information that could identify the Subject.

Randomization of the premolars or molars, which will be numbered using the Universal Numbering System (premolars = 4-5, 12-13, 20-21, or 28-29; molars = 1-3, 14-16, 17-19, or 30-32), to study treatments will be centralized and electronic. Either two pre-molars or two molars from each Subject will be randomized in a 1:1 ratio such that one of the teeth will be randomized to undergo restoration using SBU+ Adhesive (Treatment), and the other tooth will undergo restoration using SBU Adhesive (Control). Study material will be assigned according to the randomization schedule beginning with the lower tooth number in the pair.

#### 6.4.6 Intra-oral photographs

Intra-oral photographs will be taken in accordance with the Investigator's standard practice. On the day of restorations, the mouth region(s) containing the study teeth will be photographed before teeth preparation and at baseline immediately after the restoration is finished and polished. For the 6-month, 1-year, and 2-year follow-up visits, photographs will be taken before clinical performance assessments are initiated.

#### 6.4.7 Restoration and Application of Study Treatments

The restoration procedure for each lesion will be performed in accordance with the Investigator's standard practice, and both restorations should occur during a single visit.

#### 6.4.7.1 TOOTH PREPARATION & CAVITY CLEANING

After application of local anesthesia, the carious lesion will be accessed using a diamond bur. Carious dentin up to the affected dentin will then be removed using a bur, and further cavity cleansing can then be performed. Beveling of the cavity margin may be performed if it is deemed necessary in the opinion of the Investigator. After tooth preparation and cleansing, each tooth will be isolated (eg, using cotton rolls and suction, a dental isolation adapter such as Isovac<sup>TM</sup>, or a rubber dam). For preparations considered to be in deep dentin, a minimum

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


amount of calcium hydroxide followed by application of type III resin-modified glass ionomer cement (ie, 3M<sup>TM</sup> Vitrebond<sup>TM</sup> Plus) may be applied for pulp capping. Restorations for each tooth will be performed as described in Sections 6.4.7.2 and 6.4.7.3.

#### 6.4.7.2 TREATMENT GROUP – SCOTCHBOND™ UNIVERSAL PLUS ADHESIVE

For cavities/teeth in the Treatment arm, the SBU+ Adhesive will be applied following manufacturer's (3M<sup>TM</sup>) directions using a "self-etching" procedure. After application and polymerization of the adhesive using a calibrated Elipar<sup>TM</sup> DeepCure-S Curing Light (see Section 11), and after selection of an appropriate composite shade, 3M<sup>TM</sup> Filtek<sup>TM</sup> Universal Restorative will be placed in 2 mm increments and light-cured. After immediate occlusal adjustments, the restoration will be finished and polished in accordance with the Investigator's standard practice using the Sof-Lex<sup>TM</sup> Disks and the Sof-Lex<sup>TM</sup> Diamond Polishing System (see Section 11). Finishing and polishing should be similar for teeth in both treatment arms and across Subjects.

#### 6.4.7.3 CONTROL GROUP – SCOTCHBOND™ UNIVERSAL ADHESIVE

For cavities/teeth in the Control arm, the SBU Adhesive will be applied following manufacturer's (3M<sup>TM</sup>) directions using a "self-etching" procedure. After application and polymerization of the adhesive using a calibrated Elipar<sup>TM</sup> DeepCure-S Curing Light (see Section 11), and after selection of an appropriate composite shade, 3M<sup>TM</sup> Filtek<sup>TM</sup> Universal Restorative will be placed in 2 mm increments and light-cured. After immediate occlusal adjustments, the restoration will be finished and polished in accordance with the Investigator's standard practice using the Sof-Lex<sup>TM</sup> Disks and the Sof-Lex<sup>TM</sup> Diamond Polishing System (see Section 11). Finishing and polishing should be similar for teeth in both treatment arms and across Subjects.

#### 6.4.7.4 POST-RESTORATION INSTRUCTIONS

After completion of the restorations, the Investigator is to instruct the Subject to report any unusual or prolonged postoperative hypersensitivity for either study tooth that occurs during the first 7 days after the restorations.

#### **6.4.8** Post-Restoration Assessments

The clinical performance of the investigative device and comparator device, when used with 3M<sup>TM</sup> Filtek<sup>TM</sup> Universal Restorative, will be assessed by post-operative physical inspection (eg, using a mouth mirror, standardized explorers capable of allowing for marginal gap assessments, and standardized blades capable of allowing for approximal contact point assessment) of the restoration and surrounding tooth surface of teeth in each treatment arm of

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


the study in accordance with investigator's standard practice. Performance will be evaluated using criteria that include restorative material retention, fracture of restorative material, marginal adaptation, approximal anatomical form related to contact point, secondary caries, surface staining, marginal staining, color match and translucency, surface luster (ie, polish retention), and postoperative hypersensitivity. Scoring categories for each of these criteria is listed in Sections 6.4.8.1 to 6.4.8.10.

Baseline performance assessments for marginal adaptation (Section 6.4.8.3), approximal anatomical form (Section 6.4.8.4), surface and marginal staining (Sections 6.4.8.6 and 6.4.8.7, respectively), and surface luster (Section 6.4.8.9) can be performed upon removal of restoration-related isolation devices (eg, rubber dams or dental isolation adapters); however, baseline color match and translucency scoring (Section 6.4.8.8) should be performed a minimum of 30 minutes after removal of restoration-related isolation devices to allow for rehydration. For the subsequent follow-up visits, performance assessments (listed in Sections 6.4.8.1 to 6.4.8.10) should be performed after routine cleaning procedures, if applicable. In addition, performance assessments for follow-up visits should be performed after completing intra-oral photography (see Section 6.4.6).

If a tooth is withdrawn from the study (Section 6.5.2) because the tooth was missing/extracted, coronally fractured, or root canal filled, or the filling was replaced by a non-study dentist, then no further assessments will be scored for the withdrawn tooth. If a tooth is withdrawn from the study (Section 6.5.2) because of root fracture, cracks not affecting the restoration, or rampant caries, then final performance assessments listed in Sections 6.4.8.1 to 6.4.8.10 should be performed for that tooth on the day of withdrawal, excluding the postoperative hypersensitivity and tooth vitality assessment in the case of root fracture; no further assessments will be required for the withdrawn tooth after it is withdrawn.

#### 6.4.8.1 RETENTION OF RESTORATIVE MATERIAL

Categories for retention of restorative material will include:

- 1. No loss of restorative materials
- 2. Partial or complete loss of restorative materials

#### 6.4.8.2 FRACTURE OF RESTORATIVE MATERIAL

Scoring categories for the fracture of restorative material are defined as follows:

- 1. Excellent/very good: No fractures/cracks
- 2. Good: Small hairline cracks

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


- 3. Sufficient/Satisfactory: Two or more or larger hairline cracks and/or material chip fracture not affecting the marginal integrity or approximal contact
- 4. Unsatisfactory: Material chip fractures which damage marginal quality or approximal contacts

#### 6.4.8.3 MARGINAL ADAPTATION

Scoring categories for marginal adaptation are defined as follows:

- 1. Excellent/very good: No clinically detectable gap. Margins represent a harmonious continuation of the outline at the tooth/restoration transition
- 2. Good: Marginal integrity deviates from the ideal but could be upgraded to ideal by polishing. Small marginal chip fracture of the restoration can be eliminated by polishing and/or a localized gap is just perceptible. Sub-grading of good marginal adaptation should be applied as follows:
  - a. Marginal gap, white lines.
  - b. Small marginal fracture removable by polishing.
  - c. Slight ditching, slight step or small flashes, minor irregularities.
- 3. Sufficient/satisfactory: Leakage/discoloration is present but limited to the marginal area. Generalized marginal gap is easily perceptible based on clinical judgement and analysis of clinical photographs but cannot be modified without minor damage to the tooth or surrounding tissue and is not considered to result in long-term negative consequences for the tooth or surrounding tissue if left untreated. Presence of several small marginal fractures that are unlikely to cause long-term effects. Sub-grading should be applied as follows:
  - a. Gap not removable, no dentin exposure.
  - b. Several small marginal fractures.
  - c. Major irregularities, ditching or flashes, steps.
- 4. Unsatisfactory: Localized major gap that may result in exposure of dentine or base. Repair is necessary for prophylactic reasons. Sub-grading of unsatisfactory marginal adaptation should be applied as follows:
  - a. Major gap, dentine/base exposed.
  - b. Severe ditching or marginal fractures.
  - c. Larger irregularities or steps (repair necessary).

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


5. Poor: Generalized major gap or irregularities; or the restoration is loose but in situ. Replacement is necessary to prevent further damage or there are large fractures at the margins and loss of material is too extensive to be repaired.

#### 6.4.8.4 APPROXIMAL ANATOMICAL FORM (CONTACT POINT)

Scoring categories for contact points are defined as follows:

- 1. Excellent/very good: Normal contact point (floss or 25-µm metal blade can pass).
- 2. Good: Contact slightly too strong but no disadvantage (floss or 25-μm metal blade can only pass with pressure).
- 3. Sufficient/satisfactory: Somewhat weak contact, no indication of damage to tooth, gingiva, or periodontal structures (50-µm metal blade can pass).
- 4. Unsatisfactory: Too weak and possible damage due to food impaction (100-μm metal blade can pass).
- 5. Poor: Too weak and/or clear damage due to food impaction and/or pain/gingivitis.

#### 6.4.8.5 RECURRENT CARIES

Scoring categories for recurrent caries are defined as follows:

- 1. Excellent/very good: No secondary or primary caries
- 2. Good: Small and localized areas of demineralization
- 3. Sufficient/satisfactory: Larger areas of demineralization
- 4. Unsatisfactory: Caries with cavitation and suspected undermining caries
- 5. Poor: Deep caries or exposed dentin that is not accessible for repair of restoration

#### 6.4.8.6 SURFACE STAINING

Scoring categories for surface staining are as follows:

- 1. Excellent/very good: No surface staining
- 2. Good: Minor surface staining (under dry conditions), easily removable by polishing
- 3. Sufficient/satisfactory: Moderate surface staining that may also present on other teeth, not esthetically unacceptable
- 4. Unsatisfactory: Unacceptable surface staining on the restoration but not the tooth. Major intervention is necessary for improvement

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


5. Poor: Severe surface staining and/or subsurface staining, generalized or localized, not accessible for intervention (restoration may need replacement)

#### 6.4.8.7 MARGINAL STAINING

Scoring categories for marginal staining are as follows:

- 1. Excellent/very good: No marginal staining
- 2. Good: Minor marginal staining, easily removable by polishing
- 3. Sufficient/satisfactory: Moderate marginal staining, not esthetically unacceptable.
- 4. Unsatisfactory: Pronounced (mainly localized) marginal staining and not removable by polishing; major intervention necessary for improvement of esthetics
- 5. Poor: Deep marginal staining (generalized and/or profound), not accessible for intervention (restoration may need replacement)

#### 6.4.8.8 COLOR MATCH AND TRANSLUCENCY

Scoring categories for color matching are as follows:

- 1. Excellent/very good: Color and translucency of the restoration have a clinically excellent match with the surrounding enamel and adjacent teeth. There is no difference in shade, brightness or translucency between restoration and tooth.
- 2. Good: Minor deviations in shade and translucency
- 3. Sufficient/satisfactory: a clear deviation in color match that does not affect esthetics. Sub-grading of sufficient/satisfactory color match and translucency should be applied as follows:
  - a. more opaque
  - b. more translucent
  - c. darker
  - d. brighter
- 4. Unsatisfactory: There is a (localized) discoloration or opaqueness in the restoration affecting the appearance of the dentition, which can be corrected by repair (veneering) is possible. Sub-grading of unsatisfactory color match and translucency should be applied as follows:
  - a. too opaque
  - b. too translucent

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


- c. too dark
- d. too bright
- 5. Poor: The restoration displays an unacceptable alteration in color and/or translucency, and replacement is necessary

## 6.4.8.9 SURFACE LUSTER (POLISH RETENTION/(SURFACE GLOSS/ROUGHNESS)

Scoring categories for surface luster are as follows:

- 1. Excellent/very good: Surface luster is comparable to that of the surrounding enamel
- 2. Good: Surface is slightly dull but not noticeable from a speaking distance of 60-100 cm
- 3. Sufficient/satisfactory: Dull surface but still acceptable if the surface of the restoration is covered with a film of saliva
- 4. Unsatisfactory: Surface is rough and cannot be masked by salivary film. Some polishing is insufficient, and further intervention (eg, re-finishing or veneering) is necessary and possible
- 5. Poor: Surface is unacceptably rough and/or retains noticeable biofilm (plaque). Improvement by finishing or veneering is not feasible

#### 6.4.8.10 POSTOPERATIVE HYPERSENSITIVITY AND TOOTH VITALITY

Postoperative hypersensitivity upon exposure of the study tooth to a cold cotton pellet or a blast of cold air (as determined per site procedure) will be scored according to the following categories:

- 1. Excellent/very good: No hypersensitivity, normal vitality
- 2. Good: Minor hypersensitivity for a limited period of time, normal vitality
- 3. Sufficient/satisfactory: Clinically satisfactory with either of the following:
  - a. moderate hypersensitivity, or
  - b. delayed/mild sensitivity; no subjective complaints, no treatment needed
- 4. Unsatisfactory: Clinically unsatisfactory due to:
  - a. intense hypersensitivity, or
  - b. delayed sensitivity with minor subjective symptoms, or
  - c. no clinical detectable sensitivity



CLIN-PROT-CIP-11-050069


5. Poor: Intense, acute pulpitis or non-vital tooth

#### 6.4.9 Adverse Events and Adverse Device Effects

AEs and Adverse Device Effects (ADEs) will be collected from the time of restoration through the 24-month follow-up visit (optionally 3-years). AEs and ADEs will be reported according to Section 13.

#### 6.4.10 Prohibited Procedures and Treatments

Any dental procedure or treatment of the study teeth other than routine cleaning and the procedures described in Section 6.4.7 will be considered a protocol deviation. In addition, the use of peroxide-based tooth-bleaching agents applied to the study teeth is prohibited during the study and would be considered a protocol deviation.

#### 6.4.11 End of Study Documentation

Subjects may withdraw or be discontinued from this study at any time (Section 6.5 and 6.6.3). The Investigator may discontinue a Subject's study participation if the Investigator feels it is in the best interest of the Subject.

The following information will be documented at the End of Study:

- Last day of study participation
- Completion status Did the Subject complete the study (Yes/No)?
- Reason for study discontinuation

#### 6.5 SUBJECT WITHDRAWAL

#### 6.5.1 Reasons for Subject Withdrawal

Subjects may withdraw from participation in the study at any time upon request. In addition, the Investigator may choose to terminate the participation of a Subject from the study with or without their consent. The Investigator shall record the reason for withdrawal and discontinuation of the study in an applicable Case Report Form (CRF). These reasons include, but are not limited to:

- Study completion (all study related visit(s) are completed)
- Withdrawal by the Subject
- Withdrawal by Investigator
- Lost to follow-up

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


- Death
- Adverse events
- Noncompliance
- For any reason that may, in the opinion of the Investigator, negatively affect the safety or well-being of the Subject

#### 6.5.2 Reasons for Tooth Withdrawal

An individual study tooth may be withdrawn from the study at any time at the discretion of the Investigator to maintain subject safety. The Investigator shall record the reason for tooth withdrawal in an applicable CRF. These reasons include, but are not limited to:

- Cracked tooth
- Fractured tooth
- Missing / extracted tooth
- Replaced filling
- Root canal
- Rampant caries
- Other

#### 6.5.3 Handling of Withdrawal or Termination

Every effort should be made to complete assessments required for the primary endpoint and safety endpoints prior to a Subject withdrawal. In the event of Subject withdrawal or discontinuation prior to study completion (see Section 6.5.1), study Subjects will not be replaced. Screen failures or Subjects who withdraw prior to randomization to treatment will be replaced.

For study Subjects lost to follow-up, the Investigator shall make 3 documented attempts before confirming the Subject is lost to follow-up. If the study Subject withdraws from the study for any reason and there is an ongoing safety event, additional safety event information may need to be collected by the Investigator and shared with Sponsor.

Once the Subject withdraws from the study, all study teeth will be considered withdrawn. Upon Subject withdrawal, no further study evaluations will be performed, and no additional data will be collected. The Investigator may retain and continue to use any data collected before withdrawal.



CLIN-PROT-CIP-11-050069


If for any reason the Subject is withdrawn by the Investigator from this study, the Investigator will inform the Subject and the Sponsor.

If an individual study tooth is withdrawn from the study (see Section 6.5.2), then the remaining tooth may remain until study completion.

#### 6.6 VISIT SCHEDULE AND DESCRIPTION OF STUDY VISITS

#### 6.6.1 Point of Enrollment

Following recruitment and eligibility screening during Visit 1, a Subject will sign the Informed Consent Form (ICF). A Subject is considered enrolled in this study at time the informed consent form is signed by the Subject.

#### **6.6.2** Visits

After informed consent has been obtained, the following study procedures and assessments will be performed. All applicable data are to be recorded in the applicable CRFs.

#### 6.6.2.1 SCHEDULE OF EVENTS

A schedule of events is provided in Table 6.6.2.1-1 below:

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 
# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


## Table 6.6.2.1-1. Schedule of procedures and assessments by study visit.

| Procedure Description &<br>Visit Windows | Visit 1 Screening & Enrollment | Visit 2 Teeth Restorations & Baseline Follow-up | Visit 3<br>6-mo<br>Follow-up | Visit 4<br>1-yr<br>Follow-up | Visit 5<br>2-yr<br>Follow-up | Unscheduled |
|---|---|---|---|---|---|---|
| | Day -21 to 0 | Day 0 | (6 mos ± 14 d) | $(1 \text{ yr} \pm 30\text{d})$ | $(2 \text{ yr} \pm 45\text{d})$ | |
| Informed Consent | X | | | | | |
| Inclusion/Exclusion Criteria | X | X <sup>1</sup> | | | | |
| Demographics and Subject<br>Characteristics | X | | | | | |
| Teeth preparation | | X | | | | |
| Randomization | | X | | | | |
| Intra-oral photographs | | $X^2$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ |
| Restoration Procedure<br>Treatment Application | | X | | | | |
| Post-Restoration<br>Assessments | | X <sup>4</sup> | X | X | X | X |
| Adverse Events & Adverse<br>Device Effects | | X | X | X | X | X |
| End of Study | | | | | X | $X^5$ |

<sup>&</sup>lt;sup>1</sup>Confirm eligibility if screening visit and restoration occur on different days.

Release Date: 01/27/2022 08:22:29 AM CST

<sup>&</sup>lt;sup>2</sup> Before teeth preparation and immediately after the restoration is finished and polished.

<sup>&</sup>lt;sup>3</sup> Before clinical assessments are initiated.

<sup>&</sup>lt;sup>4</sup> All assessments except Color Match and Translucency performed after removal of tooth isolation devices. Color Match and Translucency assessment performed at least 30 minutes after tooth isolation device removal.

<sup>&</sup>lt;sup>5</sup> If the Subject is withdrawn early.

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


### 6.6.2.2 VISIT 1 (SCREENING & ENROLLMENT VISIT – STUDY DAY -21 TO 0)

The following procedures and assessments will be completed at Visit 1:

- 1. Assessment of eligibility, as described in Section 6.3.1
- 2. Informed consent, as described in Section 6.4.2
- 3. Undergo screening and dental assessment to corroborate that the patient meets all eligibility criteria described in Sections 6.3.1
- 4. Document Subject demographic and characteristics, as described in Section 6.4.3

## 6.6.2.3 VISIT 2 (RESTORATION PROCEDURES & BASELINE ASSESSMENTS – STUDY DAY 0)

The following procedures and assessments will be completed at Visit 2:

- 1. Confirmation that Subject meets eligibility criteria, if Visit 2 occurs on different day than Visit 1 (rescreen if > 21 days)
- 2. Teeth preparation, as described in Section 6.4.7.1
- 3. Randomization of teeth into treatment arms, as described in Section 6.4.5
- 4. Intra-oral photographs, as described in Section 6.4.6
- 5. Restoration procedure for each tooth, including application of the study treatments, as described in Section 6.4.7
- 6. All post-restoration assessments will be captured according to Section 6.4.8
- 7. Assessment and documentation of adverse events and adverse device effects, as described in Section 6.4.9

### 6.6.2.4 VISIT 3 (STUDY DAY -6 MONTHS $\pm 14$ DAYS)

The following procedures and assessments will be completed at Visit 4:

- 1. Intra-oral photographs, as described in Section 6.4.6
- 2. All post-restoration assessments will be captured according to Section 6.4.8
- 3. Assessment and documentation of adverse events and adverse device effects, as described in Section 6.4.9

### 6.6.2.5 VISIT 4 (STUDY DAY -1 YEAR $\pm$ 30 DAYS)

The following procedures and assessments will be completed at Visit 5:

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


- 1. Intra-oral photographs, as described in Section 6.4.6
- 2. All post-restoration assessments will be captured according to Section 6.4.8
- 3. Assessment and documentation of adverse events and adverse device effects, as described in Section 6.4.9

### 6.6.2.6 VISIT 5/FINAL VISIT (STUDY DAY -2 YEAR $\pm$ 45 DAYS)

The following procedures and assessments will be completed at Visit 6:

- 1. Intra-oral photographs, as described in Section 6.4.6
- 2. All post-restoration assessments will be captured according to Section 6.4.8
- 3. Assessment and documentation of adverse events and adverse device effects, as described in Section 6.4.9
- 4. Documentation of end of study, as described in Section 6.4.11

#### 6.6.2.7 UNSCHEDULED VISITS

The following procedures and assessments will be completed at any unplanned visits involving symptoms related to the study teeth:

- 1. Intra-oral photographs, as described in Section 6.4.6
- 2. All post-restoration assessments will be captured according to Section 6.4.8
- 3. Assessment and documentation of adverse events and adverse device effects, as described in Section 6.4.9
- 4. Documentation of end of study, as described in Section 6.4.11, if necessary

### 6.6.3 Point of Exit

For each Subject, the Investigator shall record the reason for withdrawal and discontinuation of the study in the applicable CRF, as described in Section 6.5.1. The Study Subject is considered to be exited from the study upon completion of the applicable CRF.

### 6.7 ROLE OF SPONSOR REPRESENTATION

### 6.7.1 Monitoring

Study monitoring is conducted to ensure that (i) the rights, safety, and well-being of study participants are protected, (ii) the reported study data are accurate, complete, and verifiable, and (iii) the conduct of the study is in compliance with the currently approved CIP, with good clinical practice (GCP) principles, and with applicable regulatory requirement(s). 3M, as



CLIN-PROT-CIP-11-050069


Sponsor of this clinical investigation, is responsible for study oversight and for providing the PI and study staff with training regarding the proper conduct of the clinical investigation with regard to CIP adherence and validity of the data recorded on the CRFs. 3M, has therefore assigned study monitor(s) to this clinical investigation. The progress of the clinical investigation will be monitored by:

- Periodic in-person and/or remote review of study documents
- Telephone and electronic communications with the study staff and PI
- Review of CRFs and source documents (eg, Subject records)

The study monitor(s), other authorized representatives of the Sponsor, representatives of the IRB/EC, or regulatory authorities may inspect all documents and records required to be maintained by the Investigator, including but not limited to, Subject records (office, clinic, or hospital) for the participants in this study. The clinical study site personnel will permit access to such records. The Investigator will give 3M study monitor(s) direct access to source documents that support data on the CRFs, including any electronic records. If site policies restrict access to Subjects' dental files to site personnel, the PI will designate a staff member to work with the Sponsor's monitor to verify source documents on an as needed basis. This verification will be conducted in a way that will ensure that only study-related information is examined.

### 6.7.2 Other Sponsor Oversight

In addition to study monitoring, the Sponsor, or their representatives may conduct the following tasks during this study:

- Audits of the Investigator
- Provision of technical support/product specific training for the study device

Investigator non-compliance of required study responsibilities will require Sponsor sanctions to alleviate the non-compliance, including corrective and preventative actions up to and including disqualification.

Details of clinical site monitoring are documented in a Monitoring Plan (MP). The MP describes in detail who will conduct the monitoring, at what frequency monitoring will be done, at what level of detail monitoring will be performed, and the distribution of monitoring reports.

### 7. STATISTICAL DESIGN AND ANALYSIS

A separate Statistical Analysis Plan (SAP) will not be generated for this study.

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


### 7.1 STATISTICAL HYPOTHESES

The objective is to compare the clinical effectiveness and safety between SBU+ Adhesive and the control, SBU Adhesive. Although the study is not powered to assess the differences in any of the endpoints between the two adhesives, comparisons will be made for exploratory purposes.

### 7.2 SAMPLE SIZE DETERMINATION

We estimate that 50 Subjects allocated to treatment are feasible in consideration of American Dental Association Guidelines<sup>31</sup> and previously published literature.<sup>9, 13</sup> The estimated sample size will account for 20% drop-outs or attrition to allow a minimum of 40 subjects completing the study. In addition, the sample size of 100 restorations (2 restorations per subject) will provide acceptable precision in estimating the overall restoration survival rate. Given an expected annual restoration failure rate of 3.3%<sup>32</sup>, a one-sided 95% confidence interval will produce an upper confidence limit of 7.7%, using the Wilson score method.

### 7.3 POPULATION FOR ANALYSES

The following analysis sets will be used:

- Full Analysis Set (FAS) Full Analysis Set will consist of all randomized Subjects who have post-baseline data available.
- Safety Set (SS) Safety Set includes all Subjects who receive either SBU+ Adhesive or SBU Adhesive for any length of time.

Prior to any interim or final analysis, the Subject(s) excluded from any statistical sensitivity analyses will be determined based on deviations deemed to impact the primary and/or secondary analyses. Critical deviations will include deviations related to restorations procedures (eg, not using SE mode), a missing assessment, and study visits outside the pre-defined windows. Subjects excluded from sensitivity analyses may differ for each time point and for each endpoint. Documentation of these decisions will occur prior to any interim analyses.

## 7.4 STATISTICAL ANALYSES

The analysis of all endpoints will be based on the FAS with and without imputation. Statistical sensitivity analyses will be performed on the primary and secondary endpoints excluding those subjects with critical deviations related to restoration procedures, missing endpoint of interest, or assessment occurring outside of scheduled follow-ups. The result of sensitivity analyses will be presented alongside the primary FAS findings. The analysis of the safety endpoint will be based on SS. There will not be any adjustment for multiplicity as the study is non-confirmatory. All analyses will be conducted using SAS software (release 9.4 or higher). Unless otherwise

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


specified, statistical tests will be two-sided and performed at a significance level of 5%. The corresponding p-values and 95% confidence intervals will be reported for all analyses.

### 7.4.1 Demographics and Baseline Characteristics

Subject demographics, baseline characteristics, and other relevant clinical information and treatment history will be summarized for all Subjects, and if relevant, by each treatment arm using descriptive statistics (frequency and percentage for categorical variables; n, mean, standard deviation, median, minimum and maximum for continuous variables).

### 7.4.2 Analysis of Primary Endpoints

The primary endpoints are the proportion of Subjects with partial or complete loss of the restoration materials, fracture grade, and marginal adaptation grade, based on the FDI World Dental Federation criteria, evaluated at 24 months. Descriptive statistics will be used to summarize the primary endpoints for overall and by the two adhesive products using FAS with imputed endpoints. The Wilcoxon signed-rank test and McNemar (or Cochran-Mantel-Haenszel) test will be used to compare the retention rate, fracture grade and marginal adaptation grade, as appropriate.

### 7.4.3 Analysis of Secondary Endpoints

The secondary endpoints (listed in Section 5.3.2) include the following:

- the proportion of Subjects with partial or complete loss of the restoration materials at 6 months and 12 months
- time to restoration failure (ie, time to partial or complete loss of restoration)
- fracture grade at 6 months and 12 months
- marginal adaptation grade at baseline, 6 months, and 12 months
- approximal anatomical form (contact point) grade at baseline, 6 months, 12 months, and 24 months
- incidence of recurrent caries at 6 months, 12 months, and 24 months
- marginal staining grade at baseline, 6 months, 12 months, and 24 months
- surface staining grade at baseline, 6 months, 12 months, and 24 months
- color match and translucency grade at baseline, 6 months, 12 months, and 24 months
- surface luster grade at baseline, 6 months, 12 months, and 24 months



CLIN-PROT-CIP-11-050069


• postoperative hypersensitivity and tooth vitality grade at 6 months, 12 months, and 24 months

These endpoints will be summarized using descriptive statistics. The Wilcoxon signed-rank test will be used to compare outcomes consisting of continuous data at each of the time points. McNemar (or Cochran-Mantel-Haenszel) test will be used to compare outcomes consisting of categorical data at each of the time points. Time to restoration failure is defined as the time between the restoration date and the first report of the presence of restoration failure. Censored observations will include surviving restorations at the date of last follow-up or completely random drop-outs. To account for multiple observations measured from the same Subjects and assume the underlying statistical assumptions are met, a marginal Cox model<sup>33, 34</sup> utilizing a robust sandwich covariance matrix estimate will be fitted to compare restoration retention survival time between the two adhesives.

### 7.4.4 Analysis of Safety Endpoint

The incidence of treatment-related adverse events throughout the study will be summarized using descriptive statistics per study arm.

#### 7.5 PLANNED INTERIM ANALYSES AND CRITERIA FOR CLINICAL INVESTIGATION

A full interim analysis will be conducted when the minimum number of FAS Subjects (Section 7.2) have completed the 12-month follow-up assessments. After all Subjects in the FAS have completed baseline and 6-month follow-up assessments, descriptive statistics will be generated. The result from the interim analysis will be used for generating a formal interim report. Given there is one full interim analysis, the O'Brien Fleming adjusted type I error rate of  $\alpha = 0.005$ , 0.048 for statistical significance will be used in the analyses conducted at 12 months and 24 months respectively. 35, 36

### 7.6 PROCEDURES FOR MISSING, UNUSED OR SPURIOUS DATA

Missing data will be displayed as missing, whereas Subjects whose data are not available (ie, "not reported", "N/A" or "not available") will be considered as a separate category and presented in the reports. Restoration failure will be information carried forward and will impact the calculation of retention rate at each subsequent visit, whereas all other endpoints under consideration that are missing will be imputed using the time-specific treatment mean for that endpoint.

#### 7.7 Procedures for Reporting Deviations from Statistical Plan

Any deviations from the planned statistical analyses described in the CIP will be documented in the final report.

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


### 7.8 VALIDATION PLAN

Validation of the statistical programs, output and result for interim and final analyses will be performed by an independent Biostatistician. The Biostatistician will also review the statistical section of the Clinical Study Report for completeness and correct interpretations of the analysis results and provide comments.

### 8. DATA MANAGEMENT

Data collected for this study will be analyzed and stored at 3M or by an approved supplier for use by researchers including those outside of the study. Permission to transmit, store and use data outside of the study will be included in the informed consent.

#### 8.1 DATA COLLECTION AND MANAGEMENT RESPONSIBILITIES

Data collection is the responsibility of the clinical study staff at the site under the supervision of the site Investigator. The Investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

All source documents should be completed in a neat, legible, permanent (ie, non-editable) manner to ensure accurate interpretation of data. Data recorded in the electronic case report form (eCRF) derived from source documents must be consistent with the data recorded on the source documents.

All data, including AEs and expected adverse event data, will be entered into a 21 CFR Part 11-compliant data capture system provided by the Sponsor. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate.

The Sponsor is responsible for compilation and verification of the clinical study data, retention of the clinical study database, performance of statistical analysis, and preparation of the clinical study report.

### 8.2 STUDY RECORDS RETENTION

The study participant's information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by the reviewing IRB, Institutional policies, regulatory authorities, or Sponsor requirements, as outlined in the study contract.

The Investigator is to contact the Sponsor prior to the destruction of any study records, and no records are to be destroyed without the written consent of the Sponsor. It is the responsibility of the Sponsor to inform the Investigator when these documents no longer need to be retained.

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


### 8.3 SPONSOR OVERSIGHT

The Investigator will allow access to clinical study records for periodic on-site or remote monitoring visits by a designated Sponsor representative, with the understanding that the representative is bound by professional secrecy and will not disclose the identity of any Subject or personal medical information. The representative will review eCRFs for completeness during monitoring visits and after the eCRFs are submitted; any discrepancies will be resolved with the Investigator or designee, as appropriate. The data will be entered into the clinical study database and verified for accuracy.

In addition to on-site or remote monitoring, routine review of submitted study information will be conducted by the Sponsor to ensure compliance with the CIP. Items reviewed include but are not limited to adverse events, deviations, number of withdrawn/terminated Subjects, which all may impact the completion of the study. Appropriate measures may be taken to ensure Investigator compliance with the CIP.

### 9. AMENDMENTS TO THE CIP

In the event that modifications to this CIP are necessary (eg, to protect the safety of the Subjects and/or the integrity of the data), the CIP will be amended and approved by the Sponsor. All changes will be evaluated for impact per the Sponsor's standard operating procedures (SOPs). In collaboration with the Investigator(s), the CIP modifications will then be documented and submitted for ethical and regulatory approval (as required) prior to implementation. Modifications will be considered implemented after all ethical and regulatory approvals (as required) are received and all key Sponsor personnel, Investigators, and Investigator designees, including key site staff, have been trained regarding the modified CIP.

### 10. DEVIATIONS FROM THE CIP

The Investigator is not allowed to deviate from the CIP except as specified in Section 5.6.4 of the International Standard, ISO/FDIS14155:2020(E). Briefly, deviations from the CIP to protect the rights, safety, and well-being of human subjects under emergency circumstances may proceed without prior approval of the Sponsor and the IRB; however, such deviations shall be documented and reported to the Sponsor and the IRB in accordance with IRB requirements. All deviations shall be documented on a deviation report form or appropriate CRF, and a deviation report form shall be completed for each event per individual Subject. The Investigator is responsible for reporting all deviations to the Sponsor and the reviewing IRB, per local requirements.



CLIN-PROT-CIP-11-050069


### 10.1 DEVIATION REPORTING TIMELINES

The timelines and methods for reporting the different types of deviations to the Sponsor are provided in Table 10.1-1.

Table 10.1-1: Timeline and method for reporting deviations

| Type of Deviation | Report to Sponsor | Method |
|---|---|---|
| Subject safety, rights, or welfare; OR | Within 24 hours of | Initial: Phone/Email to |
| Data integrity; OR | study staff becoming | Sponsor |
| Compromise the statistical analysis of | aware of event | Complete CRF |
| the study; OR | | |
| Lack of Informed Consent; OR | | |
| Inclusion/Exclusion | | |
| All other protocol deviations | Per protocol visits | Complete CRF |

## 11. DEVICE ACCOUNTABILITY

The device(s) under investigation and additional study-specific devices and equipment to be used in both arms of the study (listed in Table 11-1) will not be distributed to the investigational site until all agreements between the site and 3M are finalized and IRB approval has been obtained. 3M requires that Investigators maintain device accountability and security of the devices at all times. The Investigator or designee will:

- Maintain and account for devices at the Investigator site, including:
  - o the name(s) of person(s) who received, used, returned, or disposed of the device;
  - o the date of receipt, identification, and quantity of each investigational device (batch number/serial number or unique code);
  - o the expiration date of the device, if applicable.
- Keep devices in a secure storage area, accessible only to authorized individuals.
- Dispense devices only to Subjects properly enrolled in and eligible for the study, including the following:
  - Subject identification;
  - the date or dates of use;
  - o the date on which the investigational device was returned/explanted from Subject, if applicable.

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


- Return all unused investigational materials to the Sponsor at the end of the study or dispose of as agreed upon, including:
  - the date of return of unused, expired, or malfunctioning investigational devices, if applicable;
  - o the date and documentation of disposal of the investigational devices as per instructions of the Sponsor, if applicable.

The Sponsor shall have instructions in place and make packaging materials available, if applicable, for the safe return or disposal of investigational devices.

**Table 11-1: Device Information** 

| Device Name | Type of Product | Catalogue<br>Number |
|---|---|---|
| 3M <sup>TM</sup> Scotchbond <sup>TM</sup> Universal Plus | Dental Adhesive (new) | 41297 |
| 3M <sup>TM</sup> Scotchbond <sup>TM</sup> Universal | Dental Adhesive (control) | 41254 |
| 3M <sup>TM</sup> Filtek <sup>TM</sup> Universal Restorative | Filling material | 6555 (syringe)<br>6550 (capsule) |
| 3M <sup>TM</sup> Sof-Lex Diamond Polishing System | Pre-polishing and polishing | 5092 |
| 3M <sup>TM</sup> Sof-Lex Extra-Thin Contouring and Polishing Discs | Finishing and polishing | XT |
| 3M <sup>TM</sup> Vitrebond <sup>TM</sup> Plus Light Cure Glass Ionomer<br>Liner & Base | Liner | 7572 |
| 3M <sup>TM</sup> Elipar <sup>TM</sup> Deep Cure-S Curing Light | Light curing device | 76976 |
| Colgate <sup>TM</sup> Cavity Protection Toothpaste or<br>Crest <sup>TM</sup> Cavity Protection Toothpaste | Toothpaste | |

### 11.1 DEVICE LABELING

The devices under investigation will be labeled according to applicable regulations. A sample label will be retained, along with other study-related documents, at the site (eg, in the Investigator Site File).

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


### 11.2 ADDITIONAL STUDY-SPECIFIC EQUIPMENT/DEVICE(S)

Additional study-specific equipment/devices used in this study shall be maintained, calibrated (if applicable) and ensured to be functioning correctly during the study, in accordance with this study CIP or applicable site policy and regulatory requirements. The Sponsor should be notified of any anticipated or known issues with the device functionality that may impact the study conduct or outcome.

#### 12. STATEMENTS OF COMPLIANCE

### 12.1 ETHICAL CONSIDERATIONS

This study will be conducted in accordance with ethical principles founded in the Declaration of Helsinki. In addition, this clinical investigation shall be conducted in accordance with ISO-14155:2011 and future versions, US FDA 21 CFR parts 812, 50, 54, 56, and any regional or national regulations, as appropriate.

Approving IRBs will be provided all relevant study documentation in order to safeguard the rights, safety, and well-being of Subjects as mandated. The participating Investigator will obtain IRB approval of the study prior to initiation of the study at the site. The protocol, Instructions for Use, informed consent, written information given to Subjects, safety updates, and any revisions to these documents will be provided to the IRB by the Investigator.

### 12.2 PERIODIC REVIEWS

Ongoing reviews by IRB are required for the duration of the clinical study. The Investigator will comply with IRB requirements for ongoing reviews, at a minimum annually.

### 12.3 PARTICIPANT CONFIDENTIALITY

Participant confidentiality and privacy is strictly held in trust by the participating Investigators, their staff, and the Sponsor(s) and their authorized representatives. Information collected about Subjects during the study will be kept confidential and managed according to the requirements of the IRB and Health Insurance Portability and Accountability Act of 1996 (HIPAA). This confidentiality is extended to cover all clinical information relating to participants. Therefore, the Clinical Investigation Plan, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study, or the data will be released to any unauthorized third party without prior written approval of the Sponsor.

In the event that a Subject revokes authorization to collect or use Personal Health Information (PHI), the Investigator retains the ability to use all information collected prior to the revocation of Subject authorization.

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 



CLIN-PROT-CIP-11-050069


Study data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at 3M or approved supplier. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number (see Section 6.4.2). The electronic data capture system used by clinical sites and by 3M research staff will be secured and password protected. At the end of the study, all study databases will be archived at 3M.

### 12.4 CONFLICT OF INTEREST

The independence of this study from any actual or perceived influence, such as by the medical device industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct of this trial.

IRB/EC procedures should have provisions that the IRB/EC avoids any bias and conflict of interest, including proof of independent review of Sponsor-Investigator clinical investigations. The Sponsor can request that the IRB document that persons with conflict of interest or potential bias (eg, members of the investigation site team) were not part of the voting.

The Sponsor has established procedures for all Investigators to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest. The Sponsor will receive disclosures of conflict of interest from the PI prior to commencing the clinical investigation.

### 12.5 Insurance

The Sponsor shall provide clinical study-related insurance covering the reasonable and necessary costs of diagnostic, therapeutic, and medical treatment including hospitalization costs (treatment costs) for such participant injuries following the administration or use of the study device(s) in accordance with this clinical investigational plan and in accordance with the national regulations.

The Sponsor may reimburse the institution and/or study participants for treatment costs depending on who incurred such treatment costs. The Sponsor will not be responsible for paying for or reimbursing treatment costs if (i) the injury is attributable to the negligence or misconduct of any agent or employee of the institution or Investigator, or the failure of such persons to comply with a study protocol, (ii) the treatment costs are covered by the study participant's medical or hospital insurance coverage, or (iii) the treatment costs arose as a result of the treatment of normal progression of the study participant's disease or injuries resulting from

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


interventions that the study participants would have incurred had they not participated in the study.

## 13. ADVERSE EVENTS, ADVERSE DEVICE EFFECTS, AND DEVICE DEFICIENCIES

Investigators are responsible for ensuring that all safety events are recorded in the Subject record(s). Events defined in Section 13.1 will be reported to the Sponsor, as applicable, per the timelines in Section 13.3.

### 13.1 SAFETY AND EVENT REPORTING DEFINITIONS

This study utilizes the terms and definitions related to safety and event reporting listed in Table 13.1-1 below.

**Table 13.1-1: Safety Definitions** 

| Term | Definition |
|---|---|
| Adverse Event (AE) | Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device. |
| Adverse Device<br>Effect (ADE) | An adverse event related to the use of an investigational medical device. This includes any adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device. This includes any event that is a result of a user error or intentional misuse of the investigational device. |
| Serious Adverse<br>Event (SAE) | Any adverse event that: • Led to death • Led to serious deterioration in the health of the subject, that either resulted in • a life-threatening illness or injury • a permanent impairment of a body structure or a body function • in-patient or prolonged hospitalization • medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function |

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


| Term | Definition |
|---|---|
| | Led to fetal distress, fetal death or a congenital anomaly or<br>birth defect |
| Serious Adverse<br>Device Effect<br>(SADE) | An adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event |
| Unanticipated Serious Adverse Device Effect (USADE) | A serious adverse device effect, which by its nature, incidence, severity, or outcome has not been identified in the current version of the risk analysis report |
| Device Deficiency (DD) | An inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance, such as malfunctions, use errors, and inadequate labelling |
| Complaint | Any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness, or performance of a <b>device</b> after it is released for distribution |

### 13.2 CLASSIFICATION OF EVENTS

## 13.2.1 Severity Ratings

The severity ratings for events are defined in Table 13.2.1-1. The Investigator shall ensure rating of reportable events on the applicable Case Report Form.

**Table 13.2.1-1: Severity Ratings Definitions** 

| Term | Definition |
|---|---|
| Mild | An event that is easily tolerated by the subject, causing minimal discomfort, and not interfering with everyday activities |
| Moderate | An event that is sufficiently discomforting to interfere with normal everyday activities |
| Severe | An event that prevents normal everyday activities |

## 13.2.2 Relatedness to Study Treatment

Table 13.2.2-1 defines the relatedness definitions for events. The Investigator shall ensure rating of reportable events on the applicable Case Report Form.

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


**Table 13.2.2-1: Relatedness Definitions** 

| Term | Definition |
|---|---|
| Not Related | Relationship to the device or procedure can be excluded |
| Possible | Relationship with the use of the study device is weak but cannot be |
| | ruled out completely. |
| Causal | The event is associated with the study device or with the procedures |
| | beyond a reasonable doubt when: |
| | The event is a known side effect of the device |
| | The event has a temporal relationship with the study |
| | device/application procedures |
| | The event involves a body/site or organ that |
| | <ul> <li>The device or procedures are applied to;</li> </ul> |
| | <ul> <li>The device or procedures have an effect on</li> </ul> |
| | The event follows a known response pattern to the device |

### 13.3 REPORTING TIMELINES

Table 13.3-1 below indicates the reporting timelines and methods for reporting different types of AEs to the Sponsor. The Investigator shall also report Events to IRB/EC and local regulatory authorities, per local requirements. Reporting to Sponsor begins when study staff are aware of the event. For any event listed in the Table 13.3-1 below, the study Sponsor may request additional information from the Investigator, including but not limited to medical records, laboratory testing, or radiological results regarding the event.

Table 13.3-1. Methods and Times for Reporting Safety Events.

| Type of event | Report to Sponsor | Method |
|---|---|---|
| Adverse Events (AE) deemed by | | |
| the Investigator to be related to | | |
| participation in the study and | Per protocol visits | Complete CRF |
| considered to be due to the study | | |
| intervention or comparator product. | | |
| Unanticipated Adverse Device | Per protocol visits | Complete CRF |
| Effect (UADE) | Tel protocol visits | |
| Serious Adverse Event | Within 24 hours of | Initial: Phone/Email to |
| (SAE)/Serious Adverse Device | study staff becoming | Sponsor |
| Effect (SADE) | aware of event | Followed by: Complete CRF |



CLIN-PROT-CIP-11-050069


| Type of event | Report to Sponsor | Method |
|---|---|---|
| Unanticipated Serious Adverse | Within 24 hours of | Initial: Phone/Email to |
| Device Effect (USADE) | study staff becoming | Sponsor |
| | aware of event | Followed by: Complete CRF |
| Device Deficiency (DD) | Within 3 business | Complete CRF |
| | days of becoming | |
| | aware of event | |
| Product Complaints on 3M | Within 3 business | Complete CRF |
| Marketed Product | days of becoming | |
| | aware of event | |

### 13.4 DETAILS CONCERNING SAFETY RECORDING AND REPORTING REQUIREMENTS

### 13.4.1 Investigator

It is the responsibility of each participating Investigator to ensure all safety events (eg, AEs, SAEs, device effects, or DDs) are recorded in the Subject's record. The collection/reporting period for safety events will begin after the teeth of the Subject have been randomized. Investigators should assess for AEs at each visit, and study Subjects should be instructed to report any AE that they experience to the Investigator.

All AEs, regardless of perceived relationship to study product, will be documented in a timely manner and reported according to the methods and timelines in Section 13.3. In addition, the worsening of an underlying medical condition should also be recorded as an AE.

The AE description will include the nature of the experience (AE term), the start date, the end date, the severity of each sign or symptom, the seriousness of the event or experience, relationship to study treatment, the course of action taken, and the outcome of the experience. It will be indicated if the AE caused the Subject to be discontinued from the study.

Any AEs that are ongoing at the end of the study but are not safety-related should be marked as "persistent' per the study-specific CRF. Any Events which are related to safety OR are persistent and deemed related to the study device should be followed for up to an additional 30 calendar days or stabilization. Events reported by Subjects after the last study visit may be reported to the Sponsor up to 30 calendar days from the date of the last visit.

#### **13.4.2 Sponsor**

Safety oversight will be under the direction of the Dental Director(s) of 3M, which is composed of individuals with the appropriate expertise. The Dental Director(s) routinely reviews and assesses the safety data of the study. Emergency contact information for reporting SAEs or

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 



CLIN-PROT-CIP-11-050069


SADEs will be provided to the Investigator or Investigator designee, as well as the IRB, before initiating the study.

The Sponsor will conduct an evaluation of the received AEs and if an event is confirmed to be a SAE/UADE, will report the results of the evaluation to all regulatory agencies overseeing the project and to participating Investigators. If the Sponsor determines that the event presents an unreasonable risk to the study Subjects, the Sponsor will terminate all clinical studies or parts of studies presenting risk as soon as possible.

### 13.5 ANTICIPATED ADVERSE EVENTS AND ADVERSE DEVICE EFFECTS

Scotchbond™ Universal Plus Adhesive contains substances that may cause an allergic reaction by skin contact in certain individuals. To mitigate this potential adverse event, Subjects with a known allergy to acrylate will be excluded. In addition, the time of contact between the adhesive, especially uncured adhesive, and the Subject's oral soft tissue will be minimized. If prolonged contact with oral soft tissue occurs, the region will be flushed with large amounts of water.

### 14. VULNERABLE POPULATION

This study is intended to be conducted using a non-vulnerable population between the ages of 18-years old and 70-years old with no expectations of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate. In addition, the study includes only Subjects that are capable of providing informed consent. However, the study does not exclude economically/educationally disadvantaged persons. The protection of rights, well-being, and safety of vulnerable populations is the most important consideration and should take precedent over the interests of the study. In addition, the protection of rights, well-being, and safety of vulnerable populations, and ascertaining appended safeguards, are the prerogative of the IRB, and the Investigator should comply with all institutional guidelines related to vulnerable populations.

In recruitment process, the Investigator will ensure that Subject recruitment is free from pressure and will respect the Subject's expectations of privacy. Participation will be presented as a voluntary option. In addition, the screening process will contain procedures to assess the pregnancy status of females of childbearing age as well as the decisional capacity of potential study Subjects. The study will be described to all potential Subjects by the Investigator in non-technical terms, and the ICF will be written in an essentially non-technical manner to suit the solicited community. The study will be presented in a manner that permits ample time for consideration of participation, with no undue pressure related to the timing of the request.

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


Lastly, it is not anticipated that any special dental/medical care will be needed for any Subject enrolled for the study.

## 15. SUSPENSION OR PREMATURE TERMINATION OF THE CLINICAL INVESTIGATION PLAN

Both the Sponsor and the PI reserve the right to terminate the clinical investigation at any time. Should this be necessary, procedures will be arranged on an individual basis after review and consultation by both parties. If the study is terminated prematurely or suspended, study Subjects and the IRB will be informed promptly and provided with the reason(s) for the termination or suspension by the Sponsor or by the Investigator. If applicable, regulatory authorities and the personal dentist of the Subjects will also be informed. In terminating the clinical investigation, the 3M study team personnel and the PI will assure that adequate consideration is given to the protection of the Subjects' interests.

This study may be suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to all study participants, participating Investigators, IRB and regulatory authorities, and the Sponsor. If the study is prematurely terminated or suspended, the PI will promptly inform study participants, the IRB, and Sponsor and will provide the reason(s) for the termination or suspension. Study participants will be contacted, as applicable, and be informed of changes to study visit schedule.

Circumstances that may warrant termination or suspension include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants
- Demonstration of efficacy that would warrant stopping
- Insufficient compliance to Clinical Investigation Plan requirements
- Data that are not sufficiently complete and/or evaluable
- Determination that the primary endpoint has been met
- Determination of futility

Suspended studies may resume once concerns about safety, Clinical Investigation Plan compliance, and data quality are addressed, and satisfy the Sponsor, IRB/EC and regulatory authorities.

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


### **15.1.1 By Sponsor**

The Sponsor reserves the right to discontinue the clinical study for business or ethical reasons at any time, such as, but not limited to:

- Information regarding the study product causes doubt as to the benefit/risk ratio
- Changes in medical practice limit utility of the data obtained from the study
- Investigator(s) lack of compliance with the approved CIP, lack of oversight, and/or not following applicable regulatory or IRB/EC guidelines in conducting the study
- Incidence or severity of AEs indicates a potential health hazard or poses an unreasonable risk to the study participants
- Subject enrollment is unsatisfactory
- Fraud or misconduct

## 15.1.2 **By IRB**

The IRB/EC may choose to discontinue the study at the site for which they granted approval. If the IRB/EC discontinues the study, the Investigator will report a withdrawal of IRB/EC approval to the study Sponsor within five (5) working days.

#### 16. REGISTRATION AND PUBLICATION POLICY

#### 16.1 Public Registration

The Sponsor shall ensure that this study will comply with any required national registration requirements. This study will be conducted in accordance with the applicable publication and data sharing policies and regulations. A description of this study will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This website will not include information that identifies Subjects. At most, the website will include a summary of the results of the study and will be available for public review at any time.

### 16.2 Publications Resulting From Study

When applicable, attempts will be made to publish the results of the study, and a publication policy for this study will be addressed in a separate agreement between the PI and the Sponsor.

### 17. BIBLIOGRAPHY

1. Jeong, C.; Jeong, D., Must-know classifications of dental caries for the national dental hygiene boards. *Dentistry iQ* May 14th, 2016, 2016, pp 1-6.

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 

## CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


- 2. Stewart, C. A.; Finer, Y., Biostable, antidegradative and antimicrobial restorative systems based on host-biomaterials and microbial interactions. *Dent Mater* **2019**, *35* (1), 36-52.
- 3. Moraschini, V.; Fai, C. K.; Alto, R. M.; Dos Santos, G. O., Amalgam and resin composite longevity of posterior restorations: A systematic review and meta-analysis. *J Dent* **2015**, *43* (9), 1043-1050.
- 4. Opdam, N. J.; van de Sande, F. H.; Bronkhorst, E.; Cenci, M. S.; Bottenberg, P.; Pallesen, U.; Gaengler, P.; Lindberg, A.; Huysmans, M. C.; van Dijken, J. W., Longevity of posterior composite restorations: a systematic review and meta-analysis. *J Dent Res* **2014**, *93* (10), 943-9.
- 5. Kopperud, S. E.; Tveit, A. B.; Gaarden, T.; Sandvik, L.; Espelid, I., Longevity of posterior dental restorations and reasons for failure. *Eur J Oral Sci* **2012**, *120* (6), 539-48.
- 6. Opdam, N. J.; Bronkhorst, E. M.; Loomans, B. A.; Huysmans, M. C., 12-year survival of composite vs. amalgam restorations. *J Dent Res* **2010**, *89* (10), 1063-7.
- 7. De Munck, J.; Van Landuyt, K.; Peumans, M.; Poitevin, A.; Lambrechts, P.; Braem, M.; Van Meerbeek, B., A critical review of the durability of adhesion to tooth tissue: methods and results. *J Dent Res* **2005**, *84* (2), 118-32.
- 8. Baracco, B.; Perdigao, J.; Cabrera, E.; Ceballos, L., Two-year clinical performance of a low-shrinkage composite in posterior restorations. *Oper Dent* **2013**, *38* (6), 591-600.
- 9. Carvalho, A. A.; Leite, M. M.; Zago, J. K. M.; Nunes, C.; Barata, T. J. E.; Freitas, G. C.; Torres, E. M.; Lopes, L. G., Influence of different application protocols of universal adhesive system on the clinical behavior of Class I and II restorations of composite resin a randomized and double-blind controlled clinical trial. *BMC Oral Health* **2019**, *19* (1), 252.
- 10. Perdigao, J.; Dutra-Correa, M.; Anauate-Netto, C.; Castilhos, N.; Carmo, A. R.; Lewgoy, H. R.; Amore, R.; Cordeiro, H. J., Two-year clinical evaluation of self-etching adhesives in posterior restorations. *J Adhes Dent* **2009**, *11* (2), 149-59.
- 11. Sundfeld, R. H.; Scatolin, R. S.; Oliveira, F. G.; Machado, L. S.; Alexandre, R. S.; Sundefeld, M. L., One-year clinical evaluation of composite restorations in posterior teeth: effect of adhesive systems. *Oper Dent* **2012**, *37* (6), E1-8.
- 12. Vinagre, A.; Ramos, J.; Marques, F.; Chambino, A.; Messias, A.; Mata, A., Randomized clinical trial of five adhesive systems in occlusal restorations: One-year results. *Dent Mater J* **2020**, *39* (3), 397-406.
- 13. Balkaya, H.; Arslan, S.; Pala, K., A randomized, prospective clinical study evaluating effectiveness of a bulk-fill composite resin, a conventional composite resin and a reinforced glass ionomer in Class II cavities: one-year results. *J Appl Oral Sci* **2019**, *27*, e20180678.
- 14. Bayne, S. C.; Schmalz, G., Reprinting the classic article on USPHS evaluation methods for measuring the clinical research performance of restorative materials. *Clin Oral Investig* **2005**, *9* (4), 209-14.
- 15. Hickel, R.; Peschke, A.; Tyas, M.; Mjor, I.; Bayne, S.; Peters, M.; Hiller, K. A.; Randall, R.; Vanherle, G.; Heintze, S. D., FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. *Clin Oral Investig* **2010**, *14* (4), 349-66.

## CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


- 16. Canali, G. D.; Ignacio, S. A.; Rached, R. N.; Souza, E. M., One-year clinical evaluation of bulk-fill flowable vs. regular nanofilled composite in non-carious cervical lesions. *Clin Oral Investig* **2019**, *23* (2), 889-897.
- 17. Haak, R.; Hahnel, M.; Schneider, H.; Rosolowski, M.; Park, K. J.; Ziebolz, D.; Hafer, M., Clinical and OCT outcomes of a universal adhesive in a randomized clinical trial after 12 months. *J Dent* **2019**, *90*, 103200.
- 18. Lawson, N. C.; Robles, A.; Fu, C. C.; Lin, C. P.; Sawlani, K.; Burgess, J. O., Two-year clinical trial of a universal adhesive in total-etch and self-etch mode in non-carious cervical lesions. *J Dent* **2015**, *43* (10), 1229-34.
- 19. Lenzi, T. L.; Pires, C. W.; Soares, F. Z. M.; Raggio, D. P.; Ardenghi, T. M.; de Oliveira Rocha, R., Performance of Universal Adhesive in Primary Molars After Selective Removal of Carious Tissue: An 18-Month Randomized Clinical Trial. *Pediatr Dent* **2017**, *39* (5), 371-376.
- 20. Loguercio, A. D.; de Paula, E. A.; Hass, V.; Luque-Martinez, I.; Reis, A.; Perdigao, J., A new universal simplified adhesive: 36-Month randomized double-blind clinical trial. *J Dent* **2015**, *43* (9), 1083-1092.
- 21. Mena-Serrano, A.; Kose, C.; De Paula, E. A.; Tay, L. Y.; Reis, A.; Loguercio, A. D.; Perdigao, J., A new universal simplified adhesive: 6-month clinical evaluation. *J Esthet Restor Dent* **2013**, *25* (1), 55-69.
- 22. Munoz, M. A.; Luque, I.; Hass, V.; Reis, A.; Loguercio, A. D.; Bombarda, N. H., Immediate bonding properties of universal adhesives to dentine. *J Dent* **2013**, *41* (5), 404-11.
- 23. Olegario, I. C.; Hesse, D.; Bonecker, M.; Imparato, J. C. P.; Braga, M. M.; Mendes, F. M.; Raggio, D. P., Effectiveness of conventional treatment using bulk-fill composite resin versus Atraumatic Restorative Treatments in primary and permanent dentition: a pragmatic randomized clinical trial. *BMC Oral Health* **2017**, *17*, 34.
- 24. Perdigao, J.; Ceballos, L.; Giraldez, I.; Baracco, B.; Fuentes, M. V., Effect of a hydrophobic bonding resin on the 36-month performance of a universal adhesive-a randomized clinical trial. *Clin Oral Investig* **2020**, *24* (2), 765-776.
- 25. Perdigao, J.; Kose, C.; Mena-Serrano, A. P.; De Paula, E. A.; Tay, L. Y.; Reis, A.; Loguercio, A. D., A new universal simplified adhesive: 18-month clinical evaluation. *Oper Dent* **2014**, *39* (2), 113-27.
- 26. Shinohara, M. S.; Carvalho, P. R. M.; Neves Marcon, L.; Goncalves, D. F. M.; Ramos, F. S. E.; Fagundes, T. C., Randomized clinical trial of different adhesion strategies in noncarious cervical lesion restorations: 1-year follow-up. *Quintessence Int* **2020**, *51* (5), 352-363.
- 27. Souza, M. Y.; Jurema, A. L. B.; Caneppele, T. M. F.; Bresciani, E., Six-month performance of restorations produced with the ethanol-wet-bonding technique: a randomized trial. *Braz Oral Res* **2019**, *33*, e052.
- 28. Zanatta, R. F.; Silva, T. M.; Esper, M.; Bresciani, E.; Goncalves, S.; Caneppele, T., Bonding Performance of Simplified Adhesive Systems in Noncarious Cervical Lesions at 2-year Follow-up: A Double-blind Randomized Clinical Trial. *Oper Dent* **2019**, *44* (5), 476-487.

## CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


- 29. de Paris Matos, T.; Perdigao, J.; de Paula, E.; Coppla, F.; Hass, V.; Scheffer, R. F.; Reis, A.; Loguercio, A. D., Five-year clinical evaluation of a universal adhesive: A randomized double-blind trial. *Dent Mater* **2020**.
- 30. Demirci, M.; Tuncer, S.; Yuceokur, A. A., Prevalence of caries on individual tooth surfaces and its distribution by age and gender in university clinic patients. *Eur J Dent* **2010**, *4* (3), 270-9.
- 31. Association, A. D. Tooth-Colored Restorative Materials for Posterior Teeth; 2003.
- 32. Manhart, J.; Chen, H.; Hamm, G.; Hickel, R., Buonocore Memorial Lecture. Review of the clinical survival of direct and indirect restorations in posterior teeth of the permanent dentition. *Operative Dentistry* **2004**, *29* (5), 481-508.
- 33. Lee, E. W.; Wei, L. J.; Amato, D. A.; Leurgans, S., Cox-Type Regression Analysis for Large Numbers of Small Groups of Correlated Failure Time Observations. In *Survival Analysis: State of the Art*, Kluwer Academic Publishers: 1992; pp 237-247.
- 34. Lin, D. Y., Cox regression analysis of multivariate failure time data: the marginal approach. *Stat Med* **1994**, *13* (21), 2233-47.
- 35. Geller, N. L.; Pocock, S. J., Interim analyses in randomized clinical trials: ramifications and guidelines for practitioners. *Biometrics* **1987**, *43* (1), 213-23.
- 36. Piantadosi, S., *Clinical trials: a methodologic perspective*. John Wiley and Sons: New York, 1997; p 928.

### 18. STUDY-SPECIFIC APPENDICES

| Appendix | Title |
|---|---|
| Appendix A | American Society of Anesthesiologists (ASA) Physical Status Classification |
| | System |
| Appendix B | Grace & Smales Mobility Index |
| Appendix C | ICDAS Radiographic Scoring System |
| Appendix D | Revision History |

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 

| 3M |
|------------|
| HealthCare |

CLIN-PROT-CIP-11-050069


## 18.1 APPENDIX A. AMERICAN ASSOCIATION OF ANESTHESIOLOGISTS (ASA) PHYSICAL STATUS CLASSIFICATION SYSTEM

Last approved by the ASA House of Delegates on October 15, 2014, amended October 23, 2019

| ASA PS<br>Classification | Definition | Examples, including, but not limited to: |
|---|---|---|
| ASA I | A normal healthy patient | Healthy, non-smoking, no or minimal alcohol use |
| ASA II | A patient with mild systemic disease | Mild diseases only without substantive functional limitations. Examples include (but not limited to): current smoker, social alcohol drinker, pregnancy, obesity (30 <bmi<40), controlled="" disease<="" dm="" htn,="" lung="" mild="" td="" well-=""></bmi<40),> |
| ASA III | A patient with severe systemic disease | Substantive functional limitations; One or more moderate to severe diseases. Examples include (but not limited to): poorly controlled DM or HTN, COPD, morbid obesity (BMI ≥40), active hepatitis, alcohol dependence or abuse, implanted pacemaker, moderate reduction of ejection fraction, ESRD undergoing regularly scheduled dialysis, premature infant PCA < 60 weeks, history (>3 months) of MI, CVA, TIA, or CAD/stents. |
| ASA IV | A patient with severe systemic disease that is a constant threat to life | Examples include (but not limited to): recent (<3 months) MI, CVA, TIA, or CAD/stents, ongoing cardiac ischemia or severe valve dysfunction, severe reduction of ejection fraction, sepsis, DIC, ARD or ESRD not undergoing regularly scheduled dialysis |
| ASA V | A moribund patient who is not expected to survive without the operation | Examples include (but not limited to): ruptured abdominal/thoracic aneurysm, massive trauma, intracranial bleed with mass effect, ischemic bowel in the face of significant cardiac pathology or multiple organ/system dysfunction |
| ASA VI | A declared brain-dead patient whose organs are being removed for donor purposes f "E" denotes Emergency surgery: | |

<sup>\*</sup>The addition of "E" denotes Emergency surgery:

(An emergency is defined as existing when delay in treatment of the patient would lead to a significant increase in the threat to life or body part)

# CLINICAL INVESTIGATION PLAN

CLIN-PROT-CIP-11-050069


### 18.2 APPENDIX B. GRACE AND SMALES MOBILITY INDEX

## **Grace & Smales Mobility Index:**

- Grade 0: No apparent mobility
- Grade 1: Perceptible mobility < 1 mm in buccolingual direction
- Grade 2: Mobility > 1 mm but < 2 mm buccolingually
- Grade 3: Mobility > 2 mm buccolingually or depressibility in the socket

**3M CONFIDENTIAL** Release Date: 01/27/2022 08:22:29 AM CST 



CLIN-PROT-CIP-11-050069


### 18.3 APPENDIX C. ICDAS RADIOGRAPHIC SCORING SYSTEM

| | ICDAS Radiographic scoring system | | | |
|---|---|---|---|---|
| ICCMS™ Caries Categories | 0 | No radiolucency | | No radiolucency |
| | RA:<br>Initial stages | RA 1 | | Radiolucency in the outer ½ of the enamel |
| | | RA 2 | 0 | Radiolucency in the inner 1/2 of the enamel ± EDJ (enamel-dentine junction) |
| | | RA 3 | | Radiolucency limited to the<br>outer 1/3 of dentine |
| | RB: Moderate<br>stages | RB 4 | Q | Radiolucency reaching the middle 1/3 of dentine |
| | RC:<br>Extensive<br>stages | RC 5 | | Radiolucency reaching the inner 1/3 of dentin, clinically cavitated |
| | | RC 6 | | Radiolucency into the pulp, clinically cavitated |



CLIN-PROT-CIP-11-050069


### 18.4 APPENDIX D. REVISION HISTORY

## Overall summary of changes

Version 3. Modified Marginal Gap Adaptation grading scale to eliminate probes. Added additional detail to sample size determination and analysis of primary endpoints.

| Section | Original text | Updated text |
|---|---|---|
| modified | - <b>3</b> ····· | F |
| | <ol> <li>Good: Marginal integrity deviates from the ideal but could be upgraded to ideal by polishing. Small marginal chip fracture of the restoration can be eliminated by polishing and/or a localized gap is just perceptible with a dental probe &lt; 150 μm. Subgrading of good marginal adaptation should be applied as follows:</li> <li>Marginal gap (&lt;150 μm), white lines.</li> </ol> | <ol> <li>Good: Marginal integrity deviates from the ideal but could be upgraded to ideal by polishing. Small marginal chip fracture of the restoration can be eliminated by polishing and/or a localized gap is just perceptible. Subgrading of good marginal adaptation should be applied as follows:</li> <li>a. Marginal gap, white lines.</li> <li>b</li> <li>c</li> </ol> |
| 6.4.8.3 Marginal Adaptation | <ul> <li>b</li> <li>c</li> <li>3. Sufficient/satisfactory: Leakage/discoloration is present but limited to the marginal area. Generalized marginal gap &gt;150 μm but &lt;250 μm, is easily perceptible on probing but cannot be modified without minor damage to the tooth or surrounding tissue and is not considered to result in long-term negative consequences for the tooth or surrounding tissue if left untreated. Presence of several small marginal fractures that are unlikely to cause long-term effects. Sub-grading should be applied as follows:</li> <li>a. Gap &lt; 250 μm not removable, no dentin exposure.</li> <li>b</li> <li>c</li> </ul> | 3. Sufficient/satisfactory: Leakage/discoloration is present but limited to the marginal area. Generalized marginal gap is easily perceptible based on clinical judgement and analysis of clinical photographs but cannot be modified without minor damage to the tooth or surrounding tissue and is not considered to result in long-term negative consequences for the tooth or surrounding tissue if left untreated. Presence of several small marginal fractures that are unlikely to cause long-term effects. Sub-grading should be applied as follows: a. Gap not removable, no dentin exposure. b c |



CLIN-PROT-CIP-11-050069


## Overall summary of changes

Version 3. Modified Marginal Gap Adaptation grading scale to eliminate probes. Added additional detail to sample size determination and analysis of primary endpoints.

| Section<br>modified | Original text | Updated text |
|---|---|---|
| mounted | <ul> <li>4. Unsatisfactory: Localized gap larger than 250 μm, may result in exposure of dentine or base. Repair is necessary for prophylactic reasons. Subgrading of unsatisfactory marginal adaptation should be applied as follows:</li> <li>a. Gap &gt; 250 μm or dentine/base exposed.</li> <li>b</li> <li>c</li> <li>5. Poor: Generalized gap larger than 250 μm or the restoration is loose but in situ, re-placement is necessary to prevent further damage or there are large fractures at the margins and loss of material is too extensive to be repaired.</li> </ul> | <ol> <li>Unsatisfactory: Localized major gap that may result in exposure of dentine or base. Repair is necessary for prophylactic reasons. Sub-grading of unsatisfactory marginal adaptation should be applied as follows: <ol> <li>Major gap, dentine/base exposed.</li> <li></li> <li></li> </ol> </li> <li>Poor: Generalized major gap or irregularities; or the restoration is loose but in situ. Replacement is necessary to prevent further damage or there are large fractures at the margins and loss of material is too extensive to be repaired.</li> </ol> |
| 7.2 Sample Size<br>Determination | NA | Added: In addition, the sample size of 100 restorations (2 restorations per subject) will provide acceptable precision in estimating the overall restoration survival rate. Given an expected annual restoration failure rate of 3.3% <sup>32</sup> , a one-sided 95% confidence interval will produce an upper confidence limit of 7.7%, using the Wilson score method. |
| 7.4.2 Analysis of Primary | Descriptive statistics will be used to summarize the primary endpoints for the two adhesive | Descriptive statistics will be used to summarize the primary endpoints for overall and by the two adhesive |
| Endpoints | products using FAS with imputed endpoints. | products using FAS with imputed endpoints. |